# **Statistical Analysis Plan**

**Study ID:** 214144

**Official Title of Study:** A Phase III, Multicenter, Randomized, Active Reference, Double Blind, Double-dummy Study in Japanese Female Participants to Evaluate the Efficacy and Safety of Gepotidacin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis)

**NCT ID:** NCT05630833

**Date of Document:** 02-Apr-24

**Information Type:** Statistical Analysis Plan (SAP)

### TITLE PAGE

**Protocol Title:** A Phase III, Multicenter, Randomized, Active Reference,

Double-blind, Double-dummy Study in Japanese Female

Participants to Evaluate the Efficacy and Safety of

Gepotidacin in the Treatment of Uncomplicated Urinary Tract

Infection (Acute Cystitis)

Study Number: 214144

Compound Number: GSK2140944

**Abbreviated Title:** A study to investigate the efficacy and safety with gepotidacin

in Japanese female participants with uncomplicated urinary

tract infection (acute cystitis)

**Acronym:** EAGLE-J

Sponsor Name: GlaxoSmithKline Research & Development Limited

Regulatory Agency Identifier Number(s)

**Registry** ID

Clintrials.gov NCT05630833

XBU Statistical Analysis Plan (SAP) Template v2.0 17 January 2022

Copyright 2024 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| TIT | LE PAC | GE | | | 1 |
| \/ <b>⊏</b> I | DSION | HISTORY | <b>,</b> | | 7 |
| ۷LI | KOION | TIIOTOIX | I | | |
| 1. | INTRO | DDUCTIO | N | | 11 |
| | 1.1. | | | nds and Endpoints | |
| | 1.2. | | | | |
| 2. | | | | SES | |
| | 2.1. | Multiplic | ity Adjustm | ent | 16 |
| 3. | ANAL' | YSIS SET | ΓS | | 16 |
| 4. | | | | | |
| | 4.1. | | | ions | |
| | | 4.1.1. | | Methodology | |
| | | 4.1.2. | | Definition | |
| | | 4.1.3. | | | |
| | 4.2. | | | ) Analyses | |
| | | 4.2.1. | | of Estimands | |
| | | 4.2.2. | | ytical approach | |
| | | 4.2.3. | | analyses | |
| | | | 4.2.3.1. | - , | |
| | | | 4.2.3.2. | • | |
| | | | 4.2.3.3. | <u> </u> | |
| | | | 4.2.3.4.<br>4.2.3.5. | Tipping point analysis for missing data Impact by GCP violation | |
| | 4.3. | Second | | it(s) Analyses | |
| | 4.5. | 4.3.1. | | tic Response at TOC Visit | |
| | | 4.5.1. | 4.3.1.1. | Definition of Estimands | |
| | | | | Main analytical approach | |
| | | | 4.3.1.3. | Supplementary analyses | |
| | | 4.3.2. | | utcome and Response at the TOC Visit | |
| | | 1.0.2. | | Definition of Estimand | |
| | | | 4.3.2.2. | Main analytical approach | |
| | | 4.3.3. | | ogical Outcome and Response at the TOC | |
| | | | 4.3.3.1. | Definition of Estimand | |
| | | | 4.3.3.2. | Main analytical approach | |
| | | 4.3.4. | | tic Response at the TOC Visit in MDR | |
| | | | 4.3.4.1. | Definition of Estimand | |
| | | | 4.3.4.2. | Main analytical approach | 30 |
| | | | 4.3.4.3. | Supplementary analyses | |
| | | 4.3.5. | Clinical O | utcome and Response at the TOC Visit in MDR | 32 |
| | | | 4.3.5.1. | Definition of Estimand | |
| | | | 4.3.5.2. | Main analytical approach | |
| | | | 4.3.5.3. | Supplementary analyses | 32 |
| | | 4.3.6. | | ogical Outcome and Response at the TOC Visit | |
| | | | 4.3.6.1. | Definition of Estimand | 33 |

## **CONFIDENTIAL**

| 4.3.6.2. Main analytical approach | 34<br>34<br>35<br>35 |
|---|---|
| 4.3.6.3. Supplementary analyses 4.3.7. Investigator Assessment of Clinical Response at the TOC Visit | 34<br>34<br>35<br>35 |
| <ul> <li>4.3.7. Investigator Assessment of Clinical Response at the TOC Visit</li></ul> | 34<br>34<br>35 |
| Visit | 34<br>35<br>35 |
| 4.3.7.1. Definition of Estimand | 34<br>35<br>35 |
| 4.3.7.2. Main analytical approach | 35<br>35 |
| 4.3.8. Gepotidacin plasma and urine PK concentrations | 35 |
| 4.3.8.1. Definition of Estimand | 35<br>35 |
| 4.3.8.2. Main analytical approach | 34 |
| Exploratory Endpoint(s) Analyses | |
| CC | 36 |
| CCI | |
| Safety Analyses 4.6.1. Extent of Exposure | 44 |

| | | 4.6.2. | Adverse E | vents | .45 |
|---|---|---|---|---|---|
| | | | 4.6.2.1. | Adverse Events of Special Interest | .46 |
| | | | 4.6.2.2. | COVID-19 Assessment and COVID-19 AEs | |
| | | | 4.6.2.3. | Impact of COVID-19 Pandemic on Safety | |
| | | | | Results | .49 |
| | | | 4.6.2.4. | Quantitative Screening for Identification of | |
| | | | | Potential Adverse Reaction | .49 |
| | | | 4.6.2.5. | Impact of GCP violation | .50 |
| | | 4.6.3. | Additional | Safety Assessments | |
| | | | 4.6.3.1. | Laboratory Data | |
| | | | 4.6.3.2. | Vital Signs | |
| | | | 4.6.3.3. | ECG | .52 |
| | 4.7. | Other An | alyses | | .52 |
| | | 4.7.1. | Subgroup | analyses | .52 |
| | 4.8. | Interim A | | * | |
| | | 4.8.1. | | view | |
| | 4.9. | Changes | | I Defined Analyses | |
| | | | | • | |
| 5. | SAMP | LE SIZE D | DETERMIN | ATION | .54 |
| | 5.1. | Gepotida | cin Sample | Size | . 54 |
| | | 5.1.1. | Sample Si | ze Sensitivity | . 55 |
| | | 5.1.2. | | oin Sample Size | |
| | | 5.1.3. | Proposed | Sample Size | . 56 |
| 6. | | | | TATION | |
| | 6.1. | | | opulation Analyses | |
| | | 6.1.1. | | ulation | |
| | | 6.1.2. | | Disposition | |
| | | 6.1.3. | | hic and Baseline Characteristics | |
| | | 6.1.4. | | eviations | |
| | | 6.1.5. | | Concomitant Medications | |
| | | 6.1.6. | | rvention Compliance | |
| | | 6.1.7. | Additional | Analyses Due to the COVID-19 Pandemic | .59 |
| | 6.2. | | | rivations Rule | |
| | | 6.2.1. | Efficacy | | .60 |
| | | | | Microbiological Outcome and Response | |
| | | Ī | 6.2.1.2. | Clinical Outcome and Response | |
| | | 000 | Cafah | | |
| | | 6.2.2. | • | Advance Frents of Chariel Interset | |
| | | | 6.2.2.1. | Adverse Events of Special Interest | |
| | | 000 | 6.2.2.2. | Renal impairment | |
| | | 6.2.3. | | Potential Clinical Importance | |
| | | | 6.2.3.1. | ECG | |
| | | 604 | 6.2.3.2. | Vital Signs | ۱۵. |
| | | 6.2.4. | | Microbiology and Infectious Diseases Adult | 70 |
| | | | | ables for Adverse Event Assessment | |
| | | 6 2 E | 6.2.4.1. | Laboratory Values | |
| | | 6.2.5. | | od Study Phases for Concomitant medication | |
| | | | U.∠.IJ. I. | Study Friases for Concomitant medication | . 04 |

## **CONFIDENTIAL**

| | 6.2.5.2 Treatment Emergent Flog for Adverse Events | 0.4 |
|---|---|---|
| 6.2.6. | · | |
| 6.2.7. | | |
| 6.2.8. | Multiple measurements at One Analysis Time Point | 86 |
| 6.2.9. | | |
| 6.2.10. | | |
| DEEEDENCES | | 93 |
| | 6.2.8.<br>6.2.9.<br>6.2.10.<br>6.2.11. | <ul> <li>6.2.7. Assessment Window</li> <li>6.2.8. Multiple measurements at One Analysis Time Point</li> <li>6.2.9. Handling of Partial Dates</li> <li>6.2.10. Qualifying Uropathogen Algorithm</li> <li>6.2.11. Uropathogen Phenotype Algorithm</li> <li>6.2.12. Trademarks</li> </ul> |

214144

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | PK Summary by sampling windows | 36 |
| Table 2 | AchE-I Cumulative Grade Score Scale | 47 |
| Table 3 | Criteria for Quantitative Screening for Potential ARs. | 49 |
| Table 4 | Maximum number of participants achieving therapeutic success . | 54 |
| Table 5 | Gepotidacin Consistency Thresholds for Different Observed Gepotidacin Therapeutic Response Rate in the Global Studies and the Number of Participants on the Gepotidacin arm in this study | 55 |
| Table 6 | 95% Confidence Intervals for Different Observed Therapeutic Response Rates on the Gepotidacin arm across a Range of Differences in Therapeutic Response Rate in Gepotidacin – Nitrofurantoin assuming a 3:1 randomization. | 56 |
| Table 7 | Microbiological Outcome by Baseline Qualifying Uropathogen at the On-Therapy Visit | 60 |
| Table 8 | Microbiological Outcome and Response by Baseline Qualifying Uropathogen at the Test of Cure Visit | 60 |
| Table 9 | Microbiological Outcome and Response by Baseline Qualifying Uropathogen at the Follow Up Visit | 61 |
| Table 10 | Participant-Level Microbiological Outcome and Response Definitions per Study Visit | 62 |
| Table 11 | Microbiological Outcome by New Qualifying Uropathogen at the On Therapy Visit | 62 |
| Table 12 | Microbiological Outcome by New Qualifying Uropathogen at the Test-of-Cure Visit | 62 |
| Table 13 | Microbiological Outcome by New Qualifying Uropathogen at the Follow up Visit | 63 |
| Table 14 | Clinical Signs and Symptoms Scoring System | 64 |
| Table 15 | Clinical Outcome at the On-Therapy Visit | 64 |
| Table 16 | Clinical Outcome and Response at the Test-of-Cure Visit | 65 |
| Table 17 | Clinical Outcome and Response at the Follow-up Visit | 66 |

# **VERSION HISTORY**

| SAP Version | Approval Date | Protocol Version<br>(Date) on which<br>SAP is Based | Change | Rationale |
|---|---|---|---|---|
| SAP | 28 Nov 2022 | Amendment 02<br>(07 Nov 2022) | Not Applicable | Original version |
| SAP Amendment 1 | 02 Apr 2024 | Amendment 02<br>(07 Nov 2022) | Modified the analysis populations to exclude the participants affected by GCP violation. Modified the analysis population (micro-ITT NTF-S (Global)) to align with the primary analysis population in the global studies (204989 and 212390). Added the analysis population including the participants affected by GCP violation for the supplementary analysis. (Section 4.1.1.) Added the way of | SAP was amended based on dry-run review comments impact on the analysis populations based on the GCP violation issues that occurred in one of the sites (Site ID: PPD), caused by CI other minor edits or updates based on comparison with phase 3 studies. |
| | | | handling zero cell when computing the risk difference, and out-of-stability data for microbiological urine samples. • (Section 4.2.3.3.) Changed handling of missing data to that missing data will not be imputed in this study and missing data in the global studies will be imputed. • (Section 4.2.3.3.) Modified imputation model to align with the analyses in the global studies (204989 and 212390). | |

| | | Protocol Version | | |
|---|---|---|---|---|
| SAP Version | Approval Date | (Date) on which | Change | Rationale |
| SAP Version | Approval Date | (Date) on which SAP is Based | <ul> <li>(Section 4.2.3.3. and4.2.3.4.) Removed the computation of posterior probability.</li> <li>(Section 4.2.3.5. and 4.6.2.5.) Added the supplementary analysis including the participants affected by GCP violation for transparency.</li> <li>(Section 4.3.1.3, and 4.3.4.3.) Clarified vague component of mixture prior has "weak" information.</li> <li>(Section 4.3.1.3., and 4.3.4.3.) Added displaying median and 95%Crl of the prior for each initial weight.</li> <li>(Section 4.3.7.2. and 4.4.9.2.) Changed the analysis population from micro-ITT to ITT)</li> <li>(Section 4.3.8.2.) Added way of handling not quantifiable concentration data.</li> <li>(Section 4.3.8.2.) Changed sampling window for PK summary</li> </ul> | Rationale |

| | | Protocol Version | | |
|---|---|---|---|---|
| SAP Version | Approval Date | (Date) on which | Change | Rationale |
| | | | • CCI | |
| | | | • CCI | |
| | | | • (Section 4.6.1.) | |
| | | | Clarified the | |
| | | | definition of | |
| | | | duration. | |
| | | | (Section 4.6.2.) Added the | |
| | | | specification that | |
| | | | missing grade of | |
| | | | AE will be imputed | |
| | | | as "severe". • (Section 4.6.2.1.) | |
| | | | Clarified the | |
| | | | definition of the | |
| | | | time of onset, | |
| | | | duration, and time since end of | |
| | | | treatment. | |
| | | | • (Section 4.6.2.4.) | |
| | | | Added summary of | |
| | | | AE to screen | |
| | | | potential adverse reactions. | |
| | | | • (Section 4.6.3.1.) | |
| | | | Corrected the | |
| | | | definition of | |
| | | | increasing fold in liver chemistry. | |
| | | | • (Section 6.1.2.) | |
| | | | Removed the | |
| | | | summary of the | |
| | | | participants who is | |

| SAP Version | Approval Date | Protocol Version<br>(Date) on which<br>SAP is Based | Change | Rationale |
|---|---|---|---|---|
| SAP Version | Approval Date | (Date) on which | ongoing in this study. (Section 6.1.3.) Added and clarified some parameters in summary of baseline characteristics. (Section 6.1.7.) Removed the summary of visit impact due to COVID-19. (Table 15, 16 and 17) Clarified the derivation of clinical worsening. (Section 6.2.1.4.) Clarified MIC50 and MIC90 (Section 6.2.2.1.) Updated the list of AE term to identify AESI (Section 6.2.4.1.) Clarified the derivation of DMID grading. (Section 6.2.7) Amended the | Rationale |
| | | | assessment window. (Section 6.2.9) Amended missing/partial date of AE (Section 6.2.11) Clarified the derivation of MDR | |

# 1. INTRODUCTION

The purpose of this SAP is to describe the planned analyses to be included in the CSR for Study 214144. Details of the final analyses are provided.

# 1.1. Objectives, Estimands and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To assess the consistency of therapeutic response of gepotidacin at the Test of cure (TOC) Visit (Day 10 to 13) in female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin in Japan, with that from global studies (Studies 204989 and 212390). | Therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit |
| Secondary | |
| To assess the therapeutic response of gepotidacin compared to nitrofurantoin as an active reference descriptively, at the TOC Visit, in female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Therapeutic response at the TOC Visit |
| To assess the clinical efficacy and microbiological efficacy of gepotidacin at the TOC Visit in female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin | Clinical outcome and response at the TOC Visit Microbiological outcome and response at the TOC Visit |
| To assess the therapeutic response, clinical efficacy and microbiological efficacy of gepotidacin at the TOC Visit in female participants with acute uncomplicated cystitis who have qualifying uropathogen(s) resistant to two or more specific classes of antimicrobials at Baseline | Therapeutic response at the TOC Visit Clinical outcome and response at the TOC Visit Microbiological outcome and response at the TOC Visit |
| To assess the clinical efficacy of gepotidacin at the TOC Visit in female participants with acute uncomplicated cystitis | Investigator assessment of clinical response at the TOC Visit |
| To assess the safety and tolerability of gepotidacin in female participants with acute uncomplicated cystitis To determine the plasma and urine PK | Occurrence of treatment-emergent adverse events (AEs), serious AEs (SAEs) and adverse events of special interest (AESIs) Change from baseline in clinical laboratory tests Change from baseline in electrocardiograms (ECGs) Change from baseline in vital sign measurements Gepotidacin plasma and urine concentrations |
| concentrations of gepotidacin in female participants with acute uncomplicated cystitis | |

| Objectives | Endpoints |
|-------------|-----------|
| Exploratory | |



### **Primary estimand**

The primary clinical question of interest is: Whether the therapeutic response at the TOC visit in female participants with acute uncomplicated cystitis who have qualified uropathogen(s) at Baseline that all are susceptible to nitrofurantoin in this study is consistent with that from the global studies, regardless of intervention discontinuation for any reason. Receipt of systemic antimicrobials will impact the endpoint definition (see Section 6.2.1.1 and Section 6.2.1.2).

The estimand is described by the following attributes:

- Population: Japanese and non-Japanese (from Studies 204989 and 212390) female participants with acute uncomplicated cystitis who have qualifying uropathogen(s) at Baseline that all are susceptible to nitrofurantoin.
- Treatment condition: Gepotidacin 1500 mg BID for 5 days in this study versus gepotidacin 1500 mg BID for 5 days in the global studies (Studies 204989 and 212390) regardless of adherence.

- Variable: Therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit (the detailed definitions are provided in Section 6.2.1). Microbiological success is defined as eradication (i.e., reduction) of all qualifying bacterial uropathogens recovered at baseline to <10<sup>3</sup> colony-forming units/mL (CFU/mL) as observed on quantitative urine culture without the participant receiving other systemic antimicrobials. Clinical success is defined as resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs and symptoms) without the participant receiving other systemic antimicrobials.
- Summary measure: Comparison of the proportion of Japanese participants achieving therapeutic success in this study with 10<sup>th</sup> percentile of the predicted distribution for the proportion of participants achieving therapeutic success in this study derived from the global studies (Studies 204989 and 212390)
- Intercurrent events (ICEs):
  - Study treatment discontinuation (due to any reason) treatment policy strategy (interest is in the treatment effect regardless of study treatment discontinuation)
  - Use of systemic antimicrobials composite strategy. This ICE is captured through the definitions of microbiological and clinical response (see Section 6.2.1.1 and Section 6.2.1.2)

### **Rationale for estimand**:

Interest in this study lies in whether the efficacy of gepotidacin treatment in this study is consistent with the global studies.

The clinical question of interest in this study and the global studies (Studies 204989 and 212390) lies in the treatment effect of gepotidacin regardless of whether the full course of 5 days of treatment was taken or not, which reflects how patients may be treated in clinical practice. Hence, a treatment policy strategy is appropriate for treatment withdrawal before completing 5 days of treatment. Use of other systemic antimicrobials may confound the bacterial culture results; thus, the microbiological response will be considered failure. For clinical data, the use of a systemic antimicrobial for acute uncomplicated cystitis is a sign of treatment failure and use of a systemic antimicrobial for another infection cannot be considered a success as it confounds the assessment of efficacy. Therefore, the definition of a successful therapeutic response precludes the use of other systemic antimicrobials.

Secondary estimands are provided in Section 4.3.

# 1.2. Study Design



### 2. STATISTICAL HYPOTHESES

The primary objective is to assess the "consistency" of therapeutic success rate between the gepotidacin arm in this Eagle-J study with the pooled gepotidacin arm in the two global studies (Studies 204989 and 212390). The observed proportion of participants in the gepotidacin arm at the TOC visit achieving therapeutic success in this study will be compared with the predictive distribution of the therapeutic success rate estimated from the two global studies (Studies 204989 and 212390). "Consistency" is defined as:

$$\hat{p}_a > \frac{r_{aj}^{(10\%)}}{n_{aj}}$$

, where:

 $\hat{p}_a$ : Observed proportion of participants achieving therapeutic success on gepotidacin in this study

 $n_{aj}$ : Number of participants in gepotidacin of this study

 $r_{aj}^{(10\%)}$ : The lower 10<sup>th</sup> percentile of the cumulative distribution of the prior predictive distribution derived from the global study data for the expected number of participants achieving therapeutic success out of  $n_{aj}$  participants.

Therefore,  $\frac{r_{aj}^{(10\%)}}{n_{aj}}$  is the threshold response rate that needs to be observed to meet therapeutic success, assuming the response rate is consistent with the global study response rate. The predictive distribution is defined as:

$$r_{aj} \sim \int Binomial(r_{aj}|n_{aj},p_a) \times Beta(p_a|\alpha = r_{ag},\beta = n_{ag} - r_{ag})dp_a$$

, where:

 $r_{aj}$ : The expected number of participants achieving therapeutic success in the gepotidacin arm of this study

 $r_{ag}$ : The pooled number of participants achieving therapeutic success in the gepotidacin arm across both global studies.

 $n_{ag}$ : The pooled number of participants in the gepotidacin arms across both global studies.

The two global studies (204989 and 212390) have almost the same study design and the therapeutic response would be similar as well. Therefore, the data will be simply pooled to derive the predictive distribution.

### Example:

Assuming 884 participants on the gepotidacin arm and a 76% observed therapeutic response rate in the global studies, there is an approximately 10% probability of observing <= 56 out of 81 responders in this study if the true gepotidacin response rate in this study is consistent with the response rate estimated from the global studies. Therefore, the success rule for gepotidacin is set to require a therapeutic response rate greater than 69.1% (56/81) in order to demonstrate consistency with global results in this example.

The secondary objective is to assess the difference between the therapeutic response of gepotidacin with the nitrofurantoin therapeutic response at the TOC Visit in Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin. The difference in the therapeutic response rate between gepotidacin and nitrofurantoin will be assessed descriptively.

# 2.1. Multiplicity Adjustment

No multiplicity adjustment approaches will be used.

# 3. ANALYSIS SETS

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Study Population |
| Intent-to-Treat (all participants) (ITT-ALL) | <ul> <li>All participants who were randomly assigned to study treatment in the study.</li> <li>Participants will be analyzed according to their randomized study treatment.</li> </ul> | Listing |
| Intent-to-Treat (ITT) | All participants in ITT-ALL population, except for participants from the site (Site ID: PPD violation Participants will be analyzed according to their randomized study treatment. | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Microbiological ITT (all participants) (micro-ITT-ALL) | <ul> <li>All participants randomly assigned to study treatment who receive at least 1 dose of study treatment and have a qualifying baseline uropathogen (defined in Section 6.2.10), from a quantitative bacteriological culture of a pretreatment clean-catch midstream urine specimen.</li> <li>Participants will be analyzed according to their randomized study treatment.</li> <li>Note that qualifying uropathogens include only the uropathogen species/groups [Gram-negative bacilli (e.g. <i>E. coli, K. pneumoniae, P. mirabilis</i>), S. saprophyticus, and Enterococcus spp.], defined in Section 6.2.10.</li> </ul> | • Listing |
| Microbiological ITT (micro-ITT) | All participants in micro-ITT-ALL, except for participants from the site (Site ID: PPD due to GCP violation. Participants will be analyzed according to their randomized study treatment. | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Micro-ITT NTF-S (all participants)<br>(micro-ITT-ALL NTF-S) | All participants in the micro-<br>ITT-ALL Population whose<br>baseline qualifying bacterial | Listing |

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Micro-ITT NTF-S | uropathogens that all are susceptible to nitrofurantoin (NTF-S). Broth microdilution nitrofurantoin MIC result from JMI Laboratories (if available) will take precedence over global central laboratory (GCL) nitrofurantoin MIC result for determining susceptibility to nitrofurantoin. Nitrofurantoin susceptibility interpretations will be based on the Clinical and Laboratory Standards Institute (CLSI) guidelines Participants with missing MIC susceptibility results for any qualifying uropathogens will not be included in the NTF-S subpopulation. Participants will be analyzed according to their randomized study treatment. All participants in the micro-ITT Population whose baseline qualifying bacterial uropathogens that all are susceptible to nitrofurantoin (NTF-S). Broth microdilution nitrofurantoin MIC result from JMI Laboratories (if available) will take precedence over global central laboratory (GCL) nitrofurantoin MIC result for determining susceptibility to nitrofurantoin. Nitrofurantoin susceptibility interpretations will be based on the Clinical and Laboratory Standards Institute (CLSI) guidelines Participants with missing MIC susceptibility results for any qualifying uropathogens will not be included in the NTF-S | Study Population Efficacy |
| | <ul> <li>subpopulation.</li> <li>Participants will be analyzed according to their randomized study treatment.</li> <li>Note that this population does not include the participants in the affected site by GCP violation (Site ID: PPD ).</li> </ul> | |

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Analysis Set Micro-ITT NTF-S (Global Study) | All participants from the global studies (Studies 204989 and 212390) in the micro-ITT NTF-S (IA set) Population defined in individual studies, who are not enrolled into this study but into each of the global studies. See the individual RAP for the detailed definition of this analysis population. Note: this population will be referred as non-Japanese population. Participants will be analyzed according to their randomized | NA Analyses Evaluated NA |
| Micro-ITT NTF-S (Entire) | study treatment. All participants from micro-ITT NTF-S Population and micro-ITT NTF-S (Global Study) Population. This is the primary analysis population. Participants will be analyzed according to their randomized study treatment. | Efficacy |
| Micro-ITT-ALL NTF-S (Entire) | <ul> <li>All participants from micro-<br/>ITT-ALL NTF-S Population<br/>and micro-ITT NTF-S (Global<br/>Study) Population.</li> <li>Participants will be analyzed<br/>according to their randomized<br/>study treatment.</li> </ul> | Efficacy |
| Micro-ITT MDR | All participants in the micro-ITT Population who have any qualifying baseline bacterial uropathogens that are resistant to two or more classes of antimicrobials. See the detail for MDR definition in Section 6.2.11. Participants will be analyzed according to their randomized study treatment. | • Efficacy |
| Micro-ITT MDR (Global Study) | All participants from the global studies (Studies 204989 and 212390) in the micro-ITT Population who have any qualifying baseline bacterial uropathogens that are resistant to two or more classes of antimicrobials. See the detail for MDR definition in Section 6.2.11. | Efficacy |

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | <ul> <li>Participants will be analyzed<br/>according to their randomized<br/>study treatment.</li> </ul> | |
| Micro-ITT MDR (Entire) | <ul> <li>All participants from micro-ITT MDR Population and micro-ITT MDR (Global Study) Population.</li> <li>Participants will be analyzed according to their randomized study treatment.</li> </ul> | Efficacy |
| Safety (all participants) (Safety-ALL) | <ul> <li>All randomized participants who receive at least 1 dose of study treatment.</li> <li>Participants will be analyzed according to their actual treatment received.</li> <li>Note: if a participant receives both gepotidacin and nitrofurantoin, they will be summarized within gepotidacin 1500 mg BID.</li> </ul> | Safety |
| Safety | All randomized participants in Safety-ALL population, except for the participants from the site (Site ID: PPD ) due to GCP violation. Note: if a participant receives both gepotidacin and nitrofurantoin, they will be summarized within gepotidacin 1500 mg BID. Participants will be analyzed according to their actual study treatment received. | • Safety |
| Pharmacokinetics (all participants) (PK-ALL) | All randomized participants who receive at least 1 dose of study treatment and have at least 1 non-missing plasma or urine PK concentration (Non-quantifiable [NQ] values will be considered as non-missing values). This population will be used in the assessment and characterization of plasma and urine concentrations (summary table). Note: if a participant receives both gepotidacin and nitrofurantoin, they will be listed only (i.e. not summarized within gepotidacin 1500 mg BID). Plasma and/or urine samples for participant randomized | • Listing |

| Analysis Set | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | nitrofurantoin will not be measured. | |
| Pharmacokinetic (PK) | <ul> <li>All randomized participants in PK-ALL population, except for the participants from the site (Site ID: PPD ) due to GCP violation.</li> <li>This population will be used in the assessment and characterization of plasma and urine concentrations (summary table). Note: if a participant receives both gepotidacin and nitrofurantoin, they will be listed only (i.e., not summarized within gepotidacin 1500 mg BID). Plasma and/or urine samples for participant randomized nitrofurantoin will not be</li> </ul> | • PK |
| | nitrofurantoin will not be measured. | |

### 4. STATISTICAL ANALYSES

### 4.1. General Considerations

# 4.1.1. General Methodology

Participants who prematurely withdrew from study will not be replaced.

In the case of wrong stratification assigned at the time of randomization, the analyses will be performed based on the actual stratum per data collected in the CRF.

Confidence intervals will use 95% confidence levels unless otherwise specified.

Unless otherwise specified, continuous data will be summarized using descriptive statistics: n, mean, standard deviation (std), median, minimum and maximum. Categorical data will be summarized as the number and percentage of participants in each category.

It is anticipated that patient accrual will be spread thinly across centers and summaries of data by center would unlikely be informative and will not, therefore, be provided.

For any efficacy analyses of binary outcomes for which a risk difference will be estimated, if 100% (or 0%) success rates are observed in both treatment arms then a constant of 1E-10 will be added to each zero cell in the resultant contingency table to overcome software limitations and enable determination of the risk difference and two-sided 95% CI.

Out of stability (OOS) data may be delivered for microbiological urine samples. This data will not be included in any analysis, participants with OOS data will have their microbiological response missing and will be counted under the Unable to determine category.

Susceptibility interpretations will be based on CLSI M100 with the exception of nitroxoline and cefadroxil which are based on EUCAST guidelines and faropenem which is based on [Fuchs, 1995].

### 4.1.2. Baseline Definition

For all endpoints the baseline value will be the latest pre-dose assessment with a non-missing value (or randomization date in participants who are randomized but did not receive study treatment), including those from unscheduled visits. If time is not collected, Day 1 Pre-dose assessments are assumed to be taken prior to first dose and used as baseline.

For clinical signs and symptoms assessments and microbiological assessments, all Day 1 symptom assessments and urine samples (collected for identification of uropathogens) are used as baseline regardless of if they were taken pre or post dose. Urine samples collected on Day -1 or Day 1 can be considered as baseline.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing. If baseline data is missing, then change from baseline calculations will not be performed and will be set to missing.

### 4.1.3. Strata

Participants will be randomized to a study treatment using stratification by age category (≤ 50 years, or >50 years) and acute cystitis recurrence (nonrecurrent infection or recurrent infection). In the case of a difference between the stratification assigned at the time of randomization and the data collected in the eCRF, the data collected in the eCRF will be considered actual and used unless specified.

| Stratification Value (k) | Stratification Description |
|--------------------------|-----------------------------------|
| 1 | ≤50 years, Nonrecurrent infection |
| 2 | ≤50 years, Recurrent infection |
| 3 | >50 years, Nonrecurrent infection |
| 4 | >50 years, Recurrent infection |

# 4.2. Primary Endpoint(s) Analyses

#### 4.2.1. Definition of Estimands

Refer to Section 1.1.

# 4.2.2. Main analytical approach

The primary analysis of the primary estimand will be performed using the micro-ITT NTF-S (Entire) population.

The primary endpoint is therapeutic response (combined per-participant microbiological and clinical response) at the TOC Visit. Therapeutic success refers to participants who have been deemed both a microbiological success and a clinical success (i.e., responders).

The primary treatment effect will be estimated regardless of treatment discontinuation, as per the treatment policy strategy. The ICE of use of other systemic antimicrobial therapy is captured through the definitions of microbiological and clinical response and will be counted as failures (composite strategy). If a participant experiences both ICEs of study treatment discontinuation and use of systemic antimicrobials, then a composite strategy (assigning therapeutic response as a failure) will be used from the point that the relevant systemic antimicrobial was taken.

The number and proportion of participants achieving a therapeutic success will be presented along with its 95% Exact Clopper Pearson CI at the TOC visit and compared with the threshold for consistency with the global studies (Studies 204989 and 212390). The threshold will be derived with covariate adjustment, the covariates are the combinations of age-groups and uUTI recurrence of the participants (refer to Section 4.1.3, k=1, 2, 3, 4). For this analysis, participants who do not return for the TOC Visit or have missing data due to any reason at the TOC Visit will be treated as failures.

1. Derive the prior for therapeutic success rate in each stratum in EAGLE2/3 studies based on the definition of stratification factor (combination of age-groups and uUTI recurrence per CRF in this study

$$p_k \sim Beta(r_{k,global}, n_{k,global} - r_{k,global})$$

, where  $n_{k,global}$  and  $r_{k,global}$  are the pooled number of participants and therapeutic responders who are assigned to the gepotidacin group of  $k^{th}$  stratum (k=1, 2, 3, 4) in the micro-ITT NTF-S (Global) population, respectively.

2. Derive the predictive distribution for the number of participants achieving therapeutic success in each stratum k, (k=1, 2, 3, 4)

$$r_{k,Japan} \sim \textit{Beta binomial} \left( n_{k,Japan}, \alpha = r_{k,global}, \beta = n_{k,global} - r_{k,global} \right)$$

, where  $n_{k,Japan}$  and  $r_{k,Japan}$  are the number of participants and therapeutic responders who are assigned to the gepotidacin group of  $k^{th}$  stratum in the micro-ITT NTF-S population, respectively.

- 3. Derive lower 10 percentile as a threshold using simulation
  - a. Set j = 1
  - b. Sample  $r_{k,Japan}^{(j)}$  from  $Beta\ binomial(n_{k,Japan},\alpha=r_{k,global},\beta=n_{k,global}-r_{k,global})$  for each stratum  $(k=1,\ldots,4)$

c. Calculate 
$$r_{Japan}^{(j)} = r_{1,Japan}^{(j)} + r_{2,Japan}^{(j)} + \dots + r_{4,Japan}^{(j)}$$
 and set  $j \leftarrow j+1$ 

- d. Repeat the step b and c until j = 1,000,000.
- e. Obtain the lower 10th percentile value  $\left(r_{Japan}^{(10\%)}\right)$  of  $r_{Japan}^{(j)}$
- f. Calculate the threshold as  $r_{Japan}^{(10\%)}/n_{Japan}$  where  $n_{Japan}$  is the number of participants in the gepotidacin group.

# 4.2.3. Sensitivity analyses

### 4.2.3.1. Unadjusted threshold

The predictive distribution unadjusted of stratification factor (combination of age-groups and uUTI recurrence) is:

$$r_{aj} \sim \int Binomial(r_{aj}|n_{aj},p_a) \times Beta(p_a|\alpha = r_{ag},\beta = n_{ag} - r_{ag})dp_a$$

, where:

 $r_{aj}$ : The expected number of participants achieving therapeutic success in the gepotidacin arm of this study

 $r_{ag}$ : The pooled number of participants achieving therapeutic success in the gepotidacin arm across both global studies.

 $n_{ag}$ : The pooled number of participants in the gepotidacin arms across both global studies.

The unadjusted threshold value is defined as  $r_{aj}^{(10\%)}/n_{aj}$ , where  $r_{aj}^{(10\%)}$  is the lower 10% tile of the above predictive distribution.

### 4.2.3.2. Adjustment with randomization strata

The adjusted threshold will be calculated based on the randomization stratum the participant was randomized to (instead of the actual stratum the participant should be assigned to) using the same approach as the primary analysis (Section 4.2.2)

### 4.2.3.3. Missing data in the global studies

Sensitivity analysis on the primary estimand will be done to assess the impact of missing data using the multiple imputation method in the global studies. If the entire TOC Visit, bacteriology samples or clinical signs and symptoms assessment were missing due to COVID-19 pandemic, then the missed values will be imputed under the missing at random (MAR) assumption. If the TOC bacteriology sample was taken but a result is not available for the sample for any reason then the missed values will also be imputed under the MAR assumption. All other missing data will be considered as a failure (i.e. non-responder). A conservative approach will be taken in this study where all missing data (regardless of the reason for missingness) will be imputed as therapeutic failure.

Missing microbiological response values and clinical response values (if any) in the global studies will be imputed using separate logistic regression models under the MAR assumption in the micro-ITT NTF-S (Global) Population. The imputation models for the global studies will be estimated using the data from the global studies, respectively. The missing data in each of the global studies will be imputed using the above imputation model of each individual study. Note that the imputation models will be estimated using data on the gepotidacin arm only. The variables to be included in the imputation models are:

Models for microbiological response in the global studies:

- Age ( $\leq$ =50 years, or  $\geq$ 50 years)
- Acute cystitis recurrence (nonrecurrent infection or recurrent infection) at Baseline
- Interaction term between treatment, Baseline qualifying uropathogen species/group and MIC (gepotidacin or nitrofurantoin) for randomized treatment. This is the same variable used for multiple imputation analysis in the global studies. See the details in the study material of the global studies (204989 and 212390).
- Prior visit (On-therapy Visit) microbiological outcome

Models for clinical response in the global studies:

- Age ( $\leq$ =50 years, or  $\geq$ 50 years)
- Acute cystitis recurrence (nonrecurrent infection or recurrent infection) at Baseline
- Baseline clinical signs and symptoms total score
- Prior visit (On-therapy Visit) clinical outcome
- Site (Sites with <10 participants in the micro-ITT NTF-S Population was combined prior to unblinding of the global studies)

Any subjects that had a missing value for one or more variables listed above were excluded from the relevant imputation model(s).

### Proportion of Participants achieving therapeutic success in this study

The same approach as the primary analysis will be used.

## Threshold using the data from both global studies.

The threshold = for the lower 10<sup>th</sup> percentile of the predicted therapeutic success in this study will be calculated based on the pooled data from both global studies as follows. Note that the number of replication is set to 1,000,000.

- 1. Set i = 1
- 2. Impute missing values using separate logistic models that will be estimated using the data from both global studies.
- 3. Derive the rapeutic response from the imputed values.

- 4. Sample  $r_{k,Japan}^{(j)}$  from Beta binomial  $(n_{k,Japan}, \alpha = r_{k,global}, \beta = n_{k,global} r_{k,global})$  for each stratum (k = 1, ..., 4)
  - , where  $n_{k,Japan}$  and  $r_{k,Japan}$  are the number of participants and therapeutic responders who are assigned to the gepotidacin group of  $k^{th}$  stratum in the micro-ITT NTF-S population, respectively after imputation.
- 5. Calculate  $r_{Japan}^{(j)} = r_{1,Japan}^{(j)} + r_{2,Japan}^{(j)} + \dots + r_{4,Japan}^{(j)}$
- 6.  $j \leftarrow j + 1$
- 7. Repeat step 2-8 until j = 1,000,000
- 8. Obtain the  $10^{\text{th}}$  percentile value  $\tilde{r}_{Japan}^{(10\%)}$  from  $\{r_{Japan}^{(1)}, r_{Japan}^{(2)}, ..., r_{Japan}^{(j)}\}$  and calculate the threshold as  $\tilde{r}_{Japan}^{(10\%)}/n_{Japan}$ , where  $n_{Japan}$  is the number of participants in the gepotidacin group.

# 4.2.3.4. Tipping point analysis for missing data

The observed proportion of participants achieving therapeutic success on the gepotidacin arm in this study will be calculated using the same approach as the primary analysis.

The threshold will be derived given the assumed success rate as follows. Note that the number of replications is set to 1,000,000.

- 1. Set  $p_{global}^{(i)}$  as the assumed success rate on the gepotidacin arm in the participants with missing therapeutic response of the global studies.
- 2. Set j = 1
  - i. Set k = 1
  - ii. Draw  $r_{k,global}^{j,miss}$  from a binomial distribution (size =  $n_{k,global}^{miss}$ , probability =  $p_{global}^{(i)}$ )
    - , where  $n_{k,global}^{miss}$  and  $r_{k,global}^{j,miss}$  are the number of subjects with missing therapeutic response and the number of responders out of those with missing therapeutic response, respectively.
  - iii. Draw  $r_{k,Japan}^{(j)}$  from Beta-binomial distribution ( $size = n_{k,Japan}$ ,  $\alpha = r_{k,global}^*$ ,  $\beta = n_{k,global} r_{k,global}^*$ )

 $r_{k,global}^* = r_{k,global}^{obs} + r_{k,global}^{j,miss}$ , where  $r_{k,global}^{obs}$  is the observed number of participants achieving therapeutic success on the gepotidacin arm in  $k^{th}$  stratum of the global studies.

- iv.  $k \leftarrow k + 1$
- v. Repeat step I-V until k = K
- 3. Calculate  $r_{Japan}^{(j)} = r_{1,Japan}^{(j)} + r_{2,Japan}^{(j)} + \cdots + r_{4,Japan}^{(j)}$

- 4.  $j \leftarrow j + 1$
- 5. Repeat step 2-8 until j = 1,000,000
- 6. Obtain 10th percentile  $\tilde{r}_{Japan}^{(10\%)}$  from  $\{r_{Japan}^{(1)}, r_{Japan}^{(2)}, ..., r_{Japan}^{(j)}\}$  and calculate the threshold as  $\tilde{r}_{Japan}^{(10\%)}/n_{Japan}$ , where  $n_{Japan}$  is the number of participants in the gepotidacin group.

Tipping point analysis will be done as follows.

- 1. A grid of values will be established, ranging from 0.0 to 1.00 in steps of 2.5%, establishing the assumed therapeutic success rates on the gepotidacin arm in participants with missing therapeutic response of the global studies.
- 2. For each assumed response rate,  $p_{global}^{(i)}$ , calculate the threshold through simulation steps which is shown above.

# 4.2.3.5. Impact by GCP violation

There was GCP violation in Site PPD and the participants from the site were excluded from the primary analysis. For transparency, the sensitivity analysis including those participants will be done. This analysis is based on micro-ITT-ALL NTF-S (Entire) population. The same approach as the primary analysis except for the analysis population will be done.

# 4.3. Secondary Endpoint(s) Analyses

### 4.3.1. Therapeutic Response at TOC Visit

#### 4.3.1.1. Definition of Estimands

- **Population**: Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin
- **Treatment Condition**: Gepotidacin 1500mg BID for 5 days versus nitrofurantoin 100 mg BID for 5 days, regardless of adherence.
- **Variable**: Therapeutic response at the TOC Visit (see Section 6.2.1.1 and Section 6.2.1.2)
- **Summary Measure**: Difference in proportions of participants achieving therapeutic success in the gepotidacin and nitrofurantoin treatment groups.
- Handling of Intercurrent Event:
  - Study treatment discontinuation (due to any reason) treatment policy
  - Use of systemic antimicrobials on or prior to the visit of interest composite strategy. This ICE is captured through the definitions of microbiological and clinical response (see Section 6.2.1.1 and Section 6.2.1.2)

### 4.3.1.2. Main analytical approach

This analysis is based on micro-ITT NTF-S Population.

The number and proportion of participants achieving therapeutic success will be summarized, along with the 95% Exact Clopper Pearson CI at the TOC Visit by treatment group. ICE of use of other systemic antimicrobials is captured through the defining criteria of microbiological and clinical response (Section 6.2.1.1 and Section 6.2.1.2). Participants who do not return for the TOC Visit or have missing data at the TOC Visit will be treated as failures.

The difference in proportions of participants achieving therapeutic success for gepotidacin compared to nitrofurantoin and the 95%CI of the difference will be summarized at TOC Visit. Miettinen-Nurminen (score) confidence limits of the treatment difference will be computed. The MN estimate of the common risk difference and variance is computed by combining the point estimates and variances from individual strata using MN weights. The estimate uses inverse variance stratum weights to produce MN confidence limits for the stratum risk differences. The mathematics and algorithm of MN method can be found in the SAS procedure guide under "Summary Score Estimate of the Common Risk Difference" [SAS, 2018].

### 4.3.1.3. Supplementary analyses

Bayesian dynamic borrowing will be carried out to estimate the treatment difference in the Japanese population using data from each treatment group of the global studies (Studies 204989 and 212390).

The prior distribution is a mixture distribution with 2 components, one reflecting the results from the global studies, and a vague component reflecting 'weak information' about the treatment difference [Schmidli, 2014]

Denoting the difference (gepotidacin – nitrofurantoin) as  $\Delta$ , the prior has the form:

$$f(\Delta) = w \times f_{inf}(\Delta) + (1 - w) \times f_{vag}(\Delta)$$

- $f_{inf}(\Delta) = Normal(\Delta | \hat{\mu}_g, \hat{s}_g^2)$ : informative component
- $f_{vag}(\Delta) = Normal\left(\Delta \left| -0.10, \hat{s}_g^2 / \left(\frac{1}{n_{ag}} + \frac{1}{n_{cg}}\right)\right)$ : vague component
- $w \in [0, 1]$ : fixed initial weight

, where  $\hat{\mu}_g$ ,  $\hat{s}_g^2$  are the MN estimate of the common risk difference and variance on the proportion of participants achieving therapeutic success between gepotidacin and nitrofurantoin using the pooled data of both global studies. Similarly,  $n_{ag}$  and  $n_{cg}$  are the pooled number of participants on the gepotidacin and nitrofurantoin arms in the global studies, respectively. Note that this prior will be based on micro-ITT NTF-S (Global) Population.

The prior mixture will be updated with the MN estimate of the common risk difference and variance on the proportion of participants achieving therapeutic success between gepotidacin and nitrofurantoin using the data from this study (micro-ITT NTF-S Population) to obtain the posterior mixture. The prior and posterior median of treatment difference and 95% credible interval will be presented by each initial weight (w = 0 to 1.0 by 0.05). The other set of initial weights may be explored.

# 4.3.2. Clinical Outcome and Response at the TOC Visit

#### 4.3.2.1. Definition of Estimand

- **Population**: Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin
- Treatment Condition: Gepotidacin 1500 mg BID for 5 days, regardless of adherence
- Variable: Clinical outcome and response at the TOC Visit (see Section 6.2.1.2)

### • Summary Measure:

- Proportion of participants in each outcome category in the gepotidacin arm (Clinical outcome)
- Proportion of participants achieving clinical success in the gepotidacin arm (Clinical response)

### • Handling of Intercurrent Event:

- Study treatment discontinuation (due to any reason) treatment policy
- Use of systemic antimicrobials on or prior to the visit of interest composite strategy. This ICE is captured through the definitions of clinical response (see Section 6.2.1.2)

### 4.3.2.2. Main analytical approach

This analysis is based on micro-ITT NTF-S Population.

The number and proportion of participants achieving clinical success will be summarized, along with the 95% Exact Clopper Pearson CI at the TOC Visit by treatment group. In addition, the number and proportion of participants in each outcome category will be summarized at the TOC Visit by treatment group.

The ICE of use of other systemic antimicrobials is captured through the defining criteria of clinical outcome and response (Section 6.2.1.2). Participants who do not return for the TOC Visit or have missing data at the TOC Visit will be treated as failures.

# 4.3.3. Microbiological Outcome and Response at the TOC

#### 4.3.3.1. Definition of Estimand

- **Population**: Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) at Baseline that all are susceptible to nitrofurantoin
- Treatment Condition: Gepotidacin 1500 mg BID for 5 days, regardless of adherence
- **Variable**: Microbiological outcome and response at the TOC Visit (see Section 6.2.1.1)

### • Summary Measure:

- Proportion of participants in each outcome category in the gepotidacin arm (Microbiological outcome)
- Proportion of participants achieving microbiological success in the gepotidacin arm (Microbiological response)

# • Handling of Intercurrent Event:

- Study treatment discontinuation (due to any reason) treatment policy
- Use of systemic antimicrobials prior to the visit of interest composite strategy. This ICE is captured through the definitions of microbiological response (see Section 6.2.1.1)

## 4.3.3.2. Main analytical approach

This analysis is based on micro-ITT NTF-S Population.

The number and proportion of participants achieving microbiological success will be summarized, along with the 95% Exact Clopper Pearson CI at the TOC Visit by treatment group. In addition, the number and proportion of participants in each outcome category will be summarized at the TOC Visit by treatment group.

The ICE of use of other systemic antimicrobials is captured through the defining criteria of microbiological outcome and response (Section 6.2.1.1). Participants who do not return for the TOC Visit or have missing data at the TOC Visit will be treated as failures.

# 4.3.4. Therapeutic Response at the TOC Visit in MDR

#### 4.3.4.1. Definition of Estimand

• **Population**: Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) resistance to "two or more" specific classes of antimicrobials at Baseline(see the details in Section 6.2.11)

- Treatment Condition: Gepotidacin 1500 mg BID for 5 days, regardless of adherence
- **Variable**: Therapeutic response at the TOC Visit (see Section 6.2.1.1 and Section 6.2.1.2)
- **Summary Measure:** Proportion of participants achieving therapeutic success in the gepotidacin arm
- Handling of Intercurrent Event:
  - Study treatment discontinuation (due to any reason) treatment policy
  - Use of systemic antimicrobials on or prior to the visit of interest composite strategy. This ICE is captured through the definitions of microbiological and clinical response (see Section 6.2.1.1 and Section 6.2.1.2)

# 4.3.4.2. Main analytical approach

This analysis is based on micro-ITT MDR Population.

The number and proportion of participants with therapeutic success will be presented by treatment group at the TOC Visit along with the 95% Exact Clopper Pearson CI. Participants who do not return for the TOC Visit or have missing data a t the TOC Visit will be treated as failures.

The ICE of use of other systemic antimicrobials is captured through the defining criteria of microbiological and clinical response (Section 6.2.1.1 and Section 6.2.1.2).

### 4.3.4.3. Supplementary analyses

Additional estimand is described by the following attributes:

- **Population**: Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) resistance to "two or more" specific classes of antimicrobials at Baseline
- Treatment Condition: Gepotidacin 1500 mg BID for 5 days vs Nitrofurantoin 100 mg BID for 5 days, regardless of adherence
- Variable: Therapeutic response at the TOC Visit
- **Summary Measure:** Proportion of participants achieving therapeutic success in the gepotidacin arm
- Handling of Intercurrent Event:
  - Study treatment discontinuation (due to any reason) treatment policy
  - Use of systemic antimicrobials on or prior to the visit of interest composite strategy. This ICE is captured through the definitions of microbiological and clinical response (see Section 6.2.1.1 and Section 6.2.1.2)

Bayesian dynamic borrowing will be carried out to estimate the treatment difference in MDR subgroup in the Japanese population using pooled data from each treatment group of the global studies (Studies 204989 and 212390).

The prior distribution is a mixture distribution with 2 components, one reflecting the results from the global studies, and a vague component reflecting 'weak information' about the treatment difference [Schmidli, 2014].

Denoting the difference (gepotidacin – nitrofurantoin) as  $\Delta_{MDR}$ , the prior has the form:

$$h(\Delta_{\text{MDR}}) = w \times h_{inf}(\Delta_{\text{MDR}}) + (1 - w) \times h_{vag}(\Delta_{\text{MDR}})$$

- $h_{inf}(\Delta) = Normal(\Delta | \hat{\mu}_{g,MDR}, \hat{s}_{g,MDR}^2)$ : informative component
- $\bullet \quad h_{vag}(\Delta_{\mathrm{MDR}}) = Normal\left(\Delta \left| -0.1, \hat{s}_{g,\mathrm{MDR}}^2 \middle/ \left(\frac{1}{n_{ag,\mathrm{MDR}}} + \frac{1}{n_{cg,\mathrm{MDR}}}\right)\right) : vague \; component$
- $w \in [0,1]$ : fixed initial weight

, where  $\hat{\mu}_{g,MDR}$ ,  $\hat{s}_{g,MDR}^2$  are crude estimate of the risk difference and variance on the proportion of participants achieving therapeutic success between gepotidacin and nitrofurantoin using the pooled data from MDR subgroup of both global studies. Similarly,  $n_{ag,MDR}$  and  $n_{cg,MDR}$  are the pooled number of participants on the gepotidacin and nitrofurantoin arms in MDR subgroup of the global studies, respectively. Note that this prior will be based on micro-ITT MDR (Global) Population.

The prior mixture will be updated with the risk difference and its standard deviation derived from MDR subgroup data in this study (micro-ITT MDR population). The risk difference and its standard deviation will be obtained as follows to avoid 0 cell problem.

- 1. Beta (0.5, 0.5) will be updated with  $(n_{aj,MDR}, r_{aj,MDR})$  and  $(n_{cj,MDR}, r_{cj,MDR})$ , respectively.
- 2. Mean and variance on each treatment arm,  $(\mu_{aj,MDR}, s_{aj,MDR}^2)$  and  $(\mu_{cj,MDR}, s_{cj,MDR}^2)$ , will be obtained from each posterior.
- 3. Risk difference =  $\mu_{aj,MDR} \mu_{cj,MDR}$
- 4. Standard deviation =  $\sqrt{s_{aj,MDR}^2 + s_{cj,MDR}^2}$

, where  $n_{aj,MDR}$  and  $n_{cj,MDR}$  are the number of participants on gepotidacin and nitrofurantoin arms, respectively, and  $r_{aj,MDR}$  and  $r_{cj,MDR}$  are the number of participants achieving therapeutic success on gepotidacin and nitrofurantoin arms, respectively. The prior and posterior median and 95% credible interval will be presented by each initial weight (w = 0 to 1.0 by 0.05). The other set of initial weights may be explored.

# 4.3.5. Clinical Outcome and Response at the TOC Visit in MDR

#### 4.3.5.1. Definition of Estimand

- **Population**: Japanese female participants with acute uncomplicated cystitis who have qualifying uropathogen(s) resistance to "two or more" specific classes of antimicrobials at Baseline
- Treatment Condition: Gepotidacin 1500 mg BID for 5 days, regardless of adherence
- Variable: Clinical outcome and response at the TOC Visit (see Section 6.2.1.2)

### • Summary Measure:

- Proportion of participants in each outcome category in the gepotidacin arm (Clinical outcome)
- Proportion of participants achieving clinical success in the gepotidacin arm (Clinical response)

# • Handling of Intercurrent Event:

- Study treatment discontinuation (due to any reason) treatment policy
- Use of systemic antimicrobials on or prior to the visit of interest composite strategy. This ICE is captured through the definitions of clinical response (see Section 6.2.1.2)

### 4.3.5.2. Main analytical approach

This analysis is based on micro-ITT MDR Population.

The number and proportion of participants with clinical success will be presented by treatment group at the TOC Visit along with the 95% Exact Clopper Pearson CI. In addition, the number and proportion of participants in each outcome category will be summarized by treatment group at the TOC Visit.

The ICE of use of other systemic antimicrobials is captured through the defining criteria of clinical outcome and response (Section 6.2.1.2). Participants who do not return for the TOC Visit or have missing data at the TOC Visit will be treated as failures.

### 4.3.5.3. Supplementary analyses

Additional estimand is described by the following attributes:

- **Population**: Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) resistance to "two or more" specific classes of antimicrobials at Baseline
- **Treatment Condition**: Gepotidacin 1500 mg BID for 5 days vs Nitrofurantoin 100 mg BID for 5 days, regardless of adherence

- Variable: Clinical response at the TOC Visit
- **Summary Measure:** Proportion of participants achieving clinical success in the gepotidacin arm

### • Handling of Intercurrent Event:

- Study treatment discontinuation (due to any reason) treatment policy
- Use of systemic antimicrobials on or prior to the visit of interest composite strategy. This ICE is captured through the definitions of clinical response (see Section 6.2.1.2)

The same BDB approach will be used as therapeutic response in MDR (Refer to Section 4.3.4.3).

# 4.3.6. Microbiological Outcome and Response at the TOC Visit in MDR

### 4.3.6.1. Definition of Estimand

- **Population**: Japanese female participants with acute uncomplicated cystitis who have qualifying uropathogen(s) resistance to "two or more" specific classes of antimicrobials at Baseline
- Treatment Condition: Gepotidacin 1500 mg BID for 5 days, regardless of adherence
- **Variable**: Microbiological outcome and response at the TOC Visit (see Section 6.2.1.1)

### • Summary Measure:

- Proportion of participants in each outcome category in the gepotidacin arm (Microbiological outcome)
- Proportion of participants achieving clinical success in the gepotidacin arm (Microbiological response)

### • Handling of Intercurrent Event:

- Study treatment discontinuation (due to any reason) treatment policy
- Use of systemic antimicrobials prior to the visit of interest composite strategy. This ICE is captured through the definitions of microbiological response (see Section 6.2.1.1)

### 4.3.6.2. Main analytical approach

This analysis is based on micro-ITT MDR Population.

The number and proportion of participants with microbiological success will be presented by treatment group at the TOC Visit along with the 95% Exact Clopper Pearson CI. In addition, the number and proportion of participants in each outcome category will be summarized by treatment group at the TOC Visit.

The ICE of use of other systemic antimicrobials is captured through the defining criteria of microbiological outcome and response (Section 6.2.1.1). Participants who do not return for the TOC Visit or have missing data at the TOC Visit will be treated as failures.

### 4.3.6.3. Supplementary analyses

Additional estimand is described by the following attributes:

- **Population**: Japanese female participants with acute uncomplicated cystitis with qualifying bacterial uropathogen(s) resistance to "two or more" specific classes of antimicrobials at Baseline
- Treatment Condition: Gepotidacin 1500 mg BID for 5 days vs Nitrofurantoin 100 mg BID for 5 days, regardless of adherence
- Variable: -Microbiological response at the TOC Visit
- **Summary Measure:** Proportion of participants achieving microbiological success in the gepotidacin arm
- Handling of Intercurrent Event:
  - Study treatment discontinuation (due to any reason) treatment policy
  - Use of systemic antimicrobials prior to the visit of interest composite strategy. This ICE is captured through the definitions of microbiological response (see Section 6.2.1.1)

The same BDB approach will be used as therapeutic response in MDR (Refer to Section 4.3.4.3).

# 4.3.7. Investigator Assessment of Clinical Response at the TOC Visit

### 4.3.7.1. Definition of Estimand

- **Population**: Japanese female participants with acute uncomplicated cystitis
- **Treatment Condition**: Gepotidacin 1500 mg BID for 5 days, regardless of adherence
- Variable: Investigator assessment of clinical response at the TOC Visit
- **Summary Measure:** Proportion of participants with investigator assessed clinical response of success, failure and indeterminate/missing on the gepotidacin arm
- Handling of Intercurrent Event:
  - Study treatment discontinuation (due to any reason) treatment policy
  - Use of systemic antimicrobials on or prior to the visit of interest composite strategy

## 4.3.7.2. Main analytical approach

This analysis is based on ITT Population. Below are the categories of response and response.

| Definition | Clinical Response |
|---|---|
| Sufficient resolution of acute cystitis signs and symptoms such that no additional | Clinical Success |
| systemic antimicrobial therapy is required for the current infection | |
| Participant met any one of the criteria below: | Clinical Failure |
| No apparent response to treatment (persistence or progression of any | |
| pretreatment clinical signs and symptoms) | |
| Use of additional systemic antibiotic(s) for the current infection | |
| Death related to acute cystitis prior to the visit | |
| Determination of clinical response could not be made at the visit for any of the following | Indeterminate |
| reasons: | |
| Participant was lost to follow-up and/or the clinical assessment was not | |
| undertaken | |
| Use of confounding systemic antibiotic(s) for another infection | |
| Death prior to the visit where acute cystitis was clearly noncontributory | |

The missing data at TOC visit including outside the analysis window will be handled as shown in Section 6.2.1.5.

The number and proportion of participants with investigator assessed clinical response of success, failure and indeterminate/missing at the TOC Visit by treatment group based on ITT Population. Reasons for an assessment of failure and indeterminate responses will also be summarized.

The 95% Exact Clopper Pearson CI for the proportion of participants with success will be presented as a binomial proportion for each treatment group.

# 4.3.8. Gepotidacin plasma and urine PK concentrations

#### 4.3.8.1. Definition of Estimand

- **Population**: Japanese female participants with acute uncomplicated cystitis
- Treatment Condition: Gepotidacin 1500 mg BID for 5 days, regardless of adherence
- Variable: Gepotidacin plasma and urine PK concentrations
- **Summary Measure:** Summary statistics (appropriate for each type of endpoint) in the gepotidacin arm
- Handling of Intercurrent Event:
  - Study treatment discontinuation (due to any reason) while on treatment strategy (treatment phase defined as from first dose to On-therapy Visit)
#### 4.3.8.2. Main analytical approach

The analysis is based on the PK population.

All calculations of PK concentrations will be based on actual sampling times that fall within the set PK windows described below.

Summary statistics (n, arithmetic mean, geometric mean, median, standard deviation, minimum, maximum, 95% CI of the arithmetic and geometric means and between participant coefficient of variation [%CV and %CVb]) for plasma and urine gepotidacin concentrations will be provided by the sampling windows in Table 1. If PK concentrations are not quantifiable, these values will be imputed as 0.

PK samples collected outside of the treatment phase will only be listed.

If more than one concentration data is available within the same PK window at a scheduled time point, the data closer to 12 hours post-latest dose will only be used for the summary statistics of Pre-Dose. For Post-Dose, data closer to 2 hours post-latest dose will only be used for the summary statistics.

PK concentrations will be listed based on PK (Full) population (i.e. including the participants impacted by GCP violation).

| Visit | Parameter | PK Window |
|---|---|---|
| Baseline Study Day 1 | C <sub>day1</sub> , 0-2h | Average concentration post-dose 0 to ≤ 2 hours |
| | C <sub>day1, &gt;2h</sub> | Average concentration post-dose >2 hours |
| | C <sub>day2-5</sub> , pre-dose | Average concentration pre-dose |
| On-Therapy Study Day 2 to 5 | C <sub>day2-5</sub> , 0-2h | Average concentration post-dose 0 to ≤ 2 hours |
| | <b>C</b> day2-5, >2h | Average concentration post-dose >2 hours |

Table 1 PK Summary by sampling windows

# 4.4. Exploratory Endpoint(s) Analyses



















# 4.6. Safety Analyses

The safety analyses will be based on the Safety Analysis population, unless otherwise specified.

## 4.6.1. Extent of Exposure

Exposure will be summarized by treatment group for the Safety population using the following parameters.

- Duration of treatment (days): Rounding of the last dose date/time the first dose date/time + (0.5 in days) to the nearest integer.
- Average daily dose (mg)
- Cumulative actual dose (mg)
- Compliance rate (%)

In addition, the number of participants with <80%, >=80%-<100% and 100% compliance rate will be summarized. In addition, listing will be produced for the exposure data.

Compliance rate (%) will be calculated as:

| Study intervention | Formula |
|---|---|
| Gepotidacin/gepotidacin placebo | $\frac{total\ number\ of\ tablets\ taken}{20}*100\ (\%)$ |
| Nitrofurantoin/nitrofurantoin placebo | $\frac{total\ number\ of\ capsules\ taken}{10}*100\ (\%)$ |

#### 4.6.2. Adverse Events

An adverse event (AE) is considered treatment emergent if the AE onset date/time is on or after study intervention start date/time. If time is missing, only date will be compared. All AE and SAE summaries (including AESI) will be based on Treatment emergent adverse events unless otherwise specified.

Adverse events will be coded using the standard Medical Dictionary for Regulatory Affairs (MedDRA dictionary).

An overview summary of AEs, including counts and percentages of participants will be produced with:

- Any AE
- AE by maximum grade
- Study intervention related AEs
- AEs leading to withdrawal from study
- AEs leading to permanent discontinuation of study intervention
- AEs leading to permanent discontinuation of study intervention or withdrawal from study
- Study intervention related AEs leading to permanent discontinuation of study intervention
- SAEs
- Non-serious AEs
- Study intervention related SAE
- Fatal SAEs
- SAEs leading to permanent discontinuation of study intervention
- AEs of special interest (3 types of AESI will be provided separately)

In addition to overall summary, separate summaries of AE will be produced according to the below table. Note that missing grade of AE will be imputed as "Severe".

| | Summary by PT | Summary by PT and SOC | Summary by PT, SOC and Maximum Grade |
|---|---|---|---|
| Any AEs | | Υ | Υ |
| Study intervention related AEs | | Y | Y |
| AEs leading to permanent discontinuation of study intervention | | Y | Y |
| Common (>= 1%) AEs | Υ | | |
| Serious AEs | | Υ | Υ |
| Non-serious study intervention related AEs | Y | | |
| Serious Fatal and Non-Fatal study intervention related AEs | Y | | |

Furthermore, the following summaries will be produced for disclosure purpose.

- Summary of Common (>=5%) non-serious Adverse Events by SOC and PT (Number of Subjects and Occurrences)
- Summary of SAEs by SOC and PT (Number of Subjects and Occurrences)

A study intervention-related AE is defined as an AE for which the investigator classifies the possible relationship to study intervention as "Yes". A worst-case scenario approach will be taken to handle missing relatedness data, i.e., the summary table will include events with the relationship to study intervention as 'Yes' or missing.

A study intervention-related SAE is defined as an SAE for which the investigator classifies the relationship to study intervention as "Yes". A worst-case scenario approach will be taken to handle missing data, i.e., the summary table will include events with the relationship to study intervention as 'Yes' or missing.

Common ( $\geq$ =X%) AEs are defined as AEs with  $\geq$ =X% incidence (before rounding) in any treatment group.

The following listings will be produced.

- All Adverse Events
- Serious Adverse Events and Reasons for Considering as a Serious Adverse Event.
- Subject Profile for Death

#### 4.6.2.1. Adverse Events of Special Interest

The following will be considered adverse events of special interest (AESI) for the purpose of analyses: Clostridium difficile, Cardiovascular, Gastrointestinal, and Potential Acetylcholinesterase-Inhibition AESIs. The definitions and derivations are provided for each AESI in Section 6.2.2.1.

#### **Clostridium difficile AESIs**

This will be included in the overall summary of AEs.

## **Cardiovascular and Gastrointestinal AESIs**

The number and percentage of participants with an event will be summarized by PT, SOC and maximum grade. In addition, the incidence of AEs of GI effects and time to the first occurrence will be summarized.

#### Potential Acetylcholinesterase-Inhibition AESIs

Any reported AE listed in the Section 6.2.2.1 with a start time no later than 12 hours after the latest dose administered, as evaluated by the investigator as per the DMID grading criteria provided in the protocol Section 10.12 Appendix 12: Division of Microbiology and Infectious Disease Adult Toxicity Tables for Adverse Event Assessment, will be included in the programmatic identification of a potential Acetylcholinesterase-Inhibition (AchE-I) AESI.

Cumulative grade score of potential AchE-I events will be calculated as the sum of the grade of each reported AE. This enables the number of AEs and the severity of each AE to be taken into account. The grading scale is defined in Table 2.

Table 2 AchE-I Cumulative Grade Score Scale

| Cumulative Grade: | 0 | 1 | 2 | 3 | 4 |
|-------------------------|---|--------|--------|---------|-----|
| Cumulative Grade Score: | 0 | 1 to 3 | 4 to 6 | 7 to 10 | ≥11 |

For instance, if a participant reports two AEs, one of Grade 1 and the other of Grade 3, their cumulative grade score of 4 would result in cumulative grade 2. If a participant reports no AEs, their cumulative grade score of 0 would result in cumulative grade 0. This will be calculated for All AchE-I events, non-GI AchE-I events and GI aChE-T events, however only All AchE-I events and non-GI AchE-I events will be summarized.

AchE-I AESIs and non-GI AchE-I events will be summarized by SOC, PT and maximum grade. Separate tables will summarize AchE-I AESI by number of events and unique PT. In addition, the following parameters of AchE-I events will also be summarized, and repeated for non-GI AchE-I and GI AchE-I events.

#### **Time of onset (hours):**

#### 1. Definition

Time of onset (hours) is defined as time from first dose to the start date of the first event in hours. The first event is defined as the treatment emergent AE of which start date is the earliest within each participant. If the start time of the first event is missing, 00:00 will be imputed to calculate the time of onset. Time of onset will be rounded to the nearest hour, which will be zero hour if time of onset is <30 minutes.

#### 2. Analytical approach

Time of onset will be summarised for each type of AChE-I by treatment group.

## **Time since end of treatment (hours):**

#### 1. Definition

Time since end of treatment is defined as the time from the end date of the treatment to the non-missing end date of the last event, which will be derived as follows.

- 1) For missing end date of the treatment emergent AEs, the earliest date of death and the last contact date will be imputed.
- 2) The last event will be identified as the treatment emergent AEs of the latest end date including the imputed end date per each participant. If there are more than one AEs that have the same end date but some AEs have missing end time and the other has non-missing end time, the AE with non-missing end time will be chosen as the last event.
- 3) For missing end time of the last event, 23:59 will be imputed.
- 4) Time since end of treatment will be computed as (End date/time of the last event treatment end date/time)

#### 2. Analytical approach

For participants with the positive value of time since end of treatment which was calculated from non-missing end date, the time since end of treatment will be summarised for each category of AChE-I event (if any) by treatment group.

In addition, the following numbers will be presented for each AChE-I categories by treatment group.

- 1) The number of participants with the last AChE-I event end date imputed
- 2) The number of participants who have no event of any type of AChE-I with an end date after the end of treatment

#### **Duration (days):**

#### 1. Definition

<u>Duration in days will be computed as the difference from the start date of the first</u> event to the end date of the last event (imputed end date of last event – start date of first event + 1). The first and last events defined are the same also for the time of onset and time since end of treatment, respectively.

#### 2. Analytical approach

<u>Duration will be summarised for each AChE-I categories by treatment group.</u>

AchE-I events with a start time less than or equal to 6 hours after the latest dose administered will also be flagged in the dataset.

#### 4.6.2.2. COVID-19 Assessment and COVID-19 AEs

A standardized MedDRA Query (SMQ) will be used to identify all COVID-19 AEs. COVID-19 assessments for participants with COVID-19 AEs will be summarized.

#### 4.6.2.3. Impact of COVID-19 Pandemic on Safety Results

The summary of the incident rates of AE before and after the start of the COVID-19 will not be producedsince this study starts after the beginning of the COVID-19 pandemic.

## 4.6.2.4. Quantitative Screening for Identification of Potential Adverse Reaction

Frequentist approach to screen for potential ARs will be used. Specifically, the Crowe method [Crowe, 2013] will be applied for initial screening of the large number of adverse events to generate a "short list" of potential ARs. Due to the smaller sample size than the global studies, this method is based on the HLT relative risk (incidence rate on gepotidacin arm divided by that on nitrofurantoin arm).

Screening criteria endorsed are displayed in Table 3.

Table 3 Criteria for Quantitative Screening for Potential ARs.

| Absolute Incidence in Nitrofurantoin Subjects | HLT relative risk (Gepotidacin vs<br>Nitrofurantoin) | 95% CI for HLT RR* |
|---|---|---|
| No condition | ≥1.25 | No condition |

Note that any event which has not occurred on nitrofurantoin arm but occurred on gepotidacin arm will be included in the "short list". In addition, the following AEs will automatically be included in the "short list" of potential ARs for further qualitative evaluation:

- QT Prolongation: It is a very rare serious event that has been observed in early phase gepotidacin studies and therefore needs further evaluation. It is identified using HLT "ECG investigations".
- Serious and severe adverse events: The incidence of serious and severe AEs is expected to be very low and the qualitative assessment will be applied directly to these events without going through the quantitative screening process.
- Fungal infections: It is a known AR for nitrofurantoin. It is identified using HLT "Fungal infections NEC".
- Hepatobiliary disorders: It is a known AR for nitrofurantoin. It is identified using HLT "Hepatic and hepatobiliary disorders".
- AESI specified in Section 6.2.2.1.
- AEs with PT as "Hyperhidrosis" or "Dysarthria"

A summary table of treatment emergent adverse events meeting the pre-specified quantitative screening criteria by SOC, HLTs and PTs with incidence (%) for each treatment group, RR, and the associated 95% CI will be generated.

In addition, the following outputs will be generated.

- Summary of treatment emergent adverse events by SOC, HLT and PTs by subgroups (Consistency check between subgroups: Actual Age Category, and Renal Impairment Evaluated by Baseline CrCL)
  - Actual Age Category: <18, 18-64 and >=65
  - Renal Impairment (Baseline Creatinine Clearance): Normal (>=90mL/min), Mid-Impairment (>=60 to 89 mL/min), Moderate Impairment (>= 30 to 59 mL/min), Severe Impairment (< 30mL/min), Missing</li>
- Incidence rate of treatment emergent AEs according to different attributes by HLT and treatment group (Consistency check in AE attribute: AEs related to study treatment, AEs leading to permanent discontinuation of study treatment, AE leading to dose reduction, AE leading to dose interruption /delay, SAEs related to study treatment, Fatal SAEs, and Fatal SAEs related to study treatment)
- Summary of treatment emergent AEs by HLT and Maximum Grade (Consistency check in AE attribute)
- Summary of Cumulative Incidence of Treatment Emergent Adverse Events (HLTs) by Time to First Occurrence (Temporal association). The categories of time to first occurrence are below.
  - <= 2 days, <= 3 days, <= 4 days, <= 5 days, <= 6 days, <= 7 days, <= 8 days, <= 9 days, >= 10 days

#### 4.6.2.5. Impact of GCP violation

This analysis is based on Safety-ALL population. For transparency, the number and percentage of participants experiencing any adverse events will be presented by treatment arm, SOC and PT.

## 4.6.3. Additional Safety Assessments

#### 4.6.3.1. Laboratory Data

Summaries of worst-case grade increase from baseline grade will be provided for all the lab tests that are gradable by DMID criteria (Section 6.2.4). These summaries will display the number and percentage of subjects with a maximum post-baseline grade increasing from their baseline grade. Any increase in grade from baseline will be summarized along with any increase to a maximum grade of 3 and any increase to a maximum grade of 4. Missing baseline grade will be assumed as grade 0. For laboratory tests that are graded for both low and high values, summaries will be done separately and labelled by direction, e.g., sodium will be summarized as hyponatremia and hypernatremia separately. The determination of worst case post-baseline takes into account both planned and unscheduled assessments.

For lab tests that are not gradable by DMID criteria (Section 6.2.4), summaries of worst-case changes from baseline with respect to normal range will be generated. Decreases to low, changes to normal or no changes from baseline, and increases to high will be summarized for the worst-case post-baseline. If a subject has a decrease to low and an increase to high during the same time interval, then the subject is counted in both the "Decrease to Low" categories and the "Increase to High" categories.

Separate summary tables for change from baseline in haematology, and chemistry laboratory tests will be produced. Liver function laboratory tests will be included with chemistry lab tests.

A summary of Liver Monitoring/Stopping Event Reporting will be summarized. For participants with more than one liver stopping or liver monitoring event, only data related to the earliest most severe criteria event is included in the summary.

Abnormal liver chemistry results will be summarized by increasing folds above the upper limit of normal (ULN) including tests of interest and thresholds as follows (including data at all the visit including unscheduled visits):

- ALT or AST > 3xULN and Total Bilirubin > 2xULN\*
- ALT or AST > 3xULN and ALP < 2xULN and Total Bilirubin  $\ge 2xULN$
- ALT or AST > 3xULN and Total Bilirubin > 1.5xULN
- Hepatocellular injury: (ALT/ALT ULN)/(ALP/ALP ULN)) >= 5 and ALT >= 3xULN \*\*
- ALT or AST  $\geq 20$ xULN
- ALT or AST  $\geq 10xULN$
- ALT or AST  $\geq 8xULN$
- ALT or AST  $\geq 5$ xULN
- ALT or AST  $\geq 3xULN$
- ALT  $\geq 20$ xULN
- ALT  $\geq 10$ xULN
- ALT  $\geq 8xULN$
- ALT  $\geq$  5xULN
- ALT  $\geq 3$ xULN
- AST  $\geq 20$ xULN
- AST  $\geq 10$ xULN
- AST  $\geq 8xULN$
- AST  $\geq$  5xULN
- AST  $\geq 3xULN$

- Total Bilirubin > 2xULN
- Total Bilirubin > 1.5xULN
- Total Bilirubin > 2xULN and a portion of Direct Bilirubin >= 35% on the same day
- Total Bilirubin > 1.5xULN and a portion of Direct Bilirubin >= 35% on the same day
- \*: The total Bilirubin elevation must occur on or up to 28 days after the ALT elevation
- \*\*: sign of hepatocellular injury, ALT and ALP values must occur on the same day.

Urinalysis results will be summarized using descriptive statistics. The severity of renal impairment will be evaluated and summarized according to the method in Section 6.2.2.2.

#### 4.6.3.2. Vital Signs

The number of participants with worst case vital sign results relative to potential clinical importance (PCI) criteria which are post-baseline relative to baseline will be summarised by test and category. The summary will include baseline data and worst case post-baseline, and planned visit. The baseline categories are: Low, within Range and High for PCI criteria. The change categories for PCI criteria are: To Low, To within Range or No Change, To High. The determination of worst case post-baseline takes into account both planned and unscheduled assessments. Changes in value from baseline for each vital sign will be summarized at every assessed time point. All vital sign data will be listed.

#### 4.6.3.3. ECG

The number of participants with worst case QTc values relative to potential clinical importance criteria which are post-baseline relative to baseline will be summarised. The summary will include baseline data and worst case post-baseline, and visits (i.e. On-Therapy and TOC visits). The baseline categories are: Low, within Range and High for PCI criteria. The change categories for PCI criteria are: To Low, To within Range or No Change, To High. The determination of worst case post-baseline takes into account both planned and unscheduled assessments. A summary of change from baseline in ECG values will be produced by visit.

# 4.7. Other Analyses

#### 4.7.1. Subgroup analyses

The estimands of these subgroup analyses are the same as that provided in the Section 4.3.1.1 (therapeutic response), Section 4.3.2.1 (clinical response) and Section 4.3.3.1 (microbiological response).

These analyses are based on the micro-ITT NTF-S Population. The number and proportion of participants achieving therapeutic, clinical and microbiological success at the TOC Visit will be presented by treatment arm and the following subgroup:

- Age group:  $< 65 \text{ vs} \ge 65 \text{ years}$
- Age category (<=50, >50)
- Acute cystitis recurrence
- Actual stratification combinations as above for age category and acute cystitis recurrence
- Qualifying uropathogen species/group isolated at Baseline (including phenotypic (e.g., ESBL, MDR) and genotypic subcategories), which is defined in Section 6.2.10.
- Number of Qualified Uropathogens at Baseline (only 1 qualifying uropathogen, two qualified uropathogens, one qualified plus additional any number of non-qualified uropathogens, only for therapeutic response). If the number of participants in each subgroup is >=10, the data will be summarized. Otherwise, these will be provided in the dataset.

## 4.8. Interim Analyses

No formal interim analysis is planned. Blinded review for therapeutic, clinical and microbiological response will be conducted.

## 4.8.1. Blinded review

This blinded review aims to assess if the blinded results for the response rates are far from the expected. Once approximately 30 participants in micro-ITT NTF-S Population have completed the TOC visit, the blinded review will be done using the data from those participants. If the following criterion has been met, we will consider the response rate may be more variable than planned and the mitigation will be conducted (e.g. training for sites).

This is based on the Bayesian probability and p is pooled therapeutic success rate among gepotidacin and nitrofurantoin arms. The prior for p is Beta(0.5, 0.5) and this prior will be updated with the number of participants achieving therapeutic success and the number of participants in the blinded review (i.e. approximately 30 participants).

The maximum number of participants achieving therapeutic success to trigger considering the mitigation is provided in the Table 4. For example, if we observe <= 18 participants achieving therapeutic success in 30 participants, we will consider the mitigation.

Table 4 Maximum number of participants achieving therapeutic success

| Number of Participants in blinded review | Maximum number of participants achieving |
|---|---|
| | therapeutic success |
| 25 | 15 |
| 26 | 15 |
| 27 | 16 |
| 28 | 16 |
| 29 | 17 |
| 30 | 18 |
| 31 | 18 |
| 32 | 19 |
| 33 | 19 |
| 34 | 20 |
| 35 | 21 |

## 4.9. Changes to Protocol Defined Analyses

There were changes below to the originally planned statistical analysis specified in the protocol amendment 2 (Dated: [07-NOV-2022]).

- Added the analysis populations due to GCP violation
- Amended the micro-ITT NTF-S (Global) population to align with the primary analysis population (i.e., IA set) in the global studies (204989 and 212390).
- Originally, missing data in this study was to be imputed for tipping point analysis and multiple imputation sensitivity analysis for missing data. However, a conservative approach will be taken in this study where all missing data (regardless of the reason for missingness) will be imputed as therapeutic failure. Note that the missing data in the global studies (204989 and 212390) will be imputed for tipping point analysis and multiple imputation sensitivity analysis.

#### 5. SAMPLE SIZE DETERMINATION

This study is not designed to demonstrate non-inferiority of the gepotidacin to nitrofurantoin but designed to demonstrate consistency of this study with the global studies for therapeutic response of the gepotidacin.

# 5.1. Gepotidacin Sample Size

Approximately 81 participants in the gepotidacin treatment group is considered an appropriate sample size to evaluate consistency between this study and both global studies (Studies 204989 and 212390).

Assuming 81 participants in the micro-ITT NTF-S population on gepotidacin and an observed 76% therapeutic success rate out of 884 participants in the global studies, the

therapeutic response in the gepotidacin arm in this study would need to be greater than 69.1% to declare "consistency" with the global studies.

## 5.1.1. Sample Size Sensitivity

Table 5 demonstrates a range of observed therapeutic response rates and the number of participants on the gepotidacin arm in this study against the corresponding consistency thresholds required in this study assuming 884 participants on the gepotidacin arm in both global studies.

Table 5 Gepotidacin Consistency Thresholds for Different Observed Gepotidacin Therapeutic Response Rate in the Global Studies and the Number of Participants on the Gepotidacin arm in this study

| Observed | | Number of Participants on the Gepotidacin arm in this study | | | | | |
|---|---|---|---|---|---|---|---|
| Therapeutic Response Rate in | 75 | 77 | 79 | 81 | 83 | 85 | 87 |
| the Global Studies | 07.00/ | 07.70/ | 00.00/ | 07.00/ | 07.00/ | 07.00/ | 07.00/ |
| 45% | 37.3% | 37.7% | 38.0% | 37.0% | 37.3% | 37.6% | 37.9% |
| 50% | 42.7% | 42.9% | 43.0% | 42.0% | 42.2% | 42.4% | 42.5% |
| 55% | 46.7% | 46.8% | 48.1% | 48.1% | 48.2% | 48.2% | 48.3% |
| 60% | 52.0% | 51.9% | 53.2% | 53.1% | 53.0% | 52.9% | 52.9% |
| 65% | 57.3% | 57.1% | 58.2% | 58.0% | 57.8% | 57.6% | 58.6% |
| 70% | 62.7% | 63.6% | 63.3% | 63.0% | 62.7% | 63.5% | 63.2% |
| 75% | 68.0% | 68.8% | 68.4% | 67.9% | 68.7% | 68.2% | 69.0% |
| 80% | 73.3% | 74.0% | 73.4% | 74.1% | 73.5% | 74.1% | 74.7% |

## 5.1.2. Nitrofurantoin Sample Size

The sample size on the nitrofurantoin arm is based on the precision estimate of 95%CI for the treatment difference.

The treatment difference between gepotidacin and nitrofurantoin will be assessed descriptively. Table 6 demonstrates a range of observed differences and corresponding 95% CIs assuming a 3:1 randomization (i.e. 81 participants on gepotidacin and 27 on nitrofurantoin in micro-ITT NTF-S population).

Table 6 95% Confidence Intervals for Different Observed Therapeutic Response Rates on the Gepotidacin arm across a Range of Differences in Therapeutic Response Rate in Gepotidacin – Nitrofurantoin assuming a 3:1 randomization.

| Observed Gepo | Observed difference of TRR in Gepotidacin from that in Nitrofurantoin and corresponding | | | | |
|---|---|---|---|---|---|
| TRR | | | 95% CI (%) | | |
| | 10% | 5% | 0% | -5% | -10% |
| 45% | (-11.0,31.0) | (-16.4,26.4) | (-21.7,21.7) | (-26.8,16.8) | (-31.7,11.7) |
| 50% | (-11.4,31.4) | (-16.7,26.7) | (-21.8,21.8) | (-26.7,16.7) | (-31.4,11.4) |
| 55% | (-11.7,31.7) | (-16.8,26.8) | (-21.7,21.7) | (-26.4,16.4) | (-31.0,11.0) |
| 60% | (-11.7,31.7) | (-16.6,26.6) | (-21.3,21.3) | (-25.9,15.9) | (-30.3,10.3) |
| 65% | (-11.4,31.4) | (-16.2,26.2) | (-20.8,20.8) | (-25.2,15.2) | (-29.4,9.4) |
| 70% | (-11.0,31.0) | (-15.6,25.6) | (-20.0,20.0) | (-24.1,14.1) | (-28.1,8.1) |
| 75% | (-10.3,30.3) | (-14.7,24.7) | (-18.9,18.9) | (-22.8,12.8) | (-26.4,6.4) |
| 80% | (-9.4,29.4) | (-13.5,23.5) | (-17.4,17.4) | (-21.0,11.0) | (-24.3,4.3) |

## 5.1.3. Proposed Sample Size

Assuming a 36% evaluability rate, approximately 300 participants will be enrolled and randomized to either gepotidacin or nitrofurantoin in a 3:1 ratio to achieve 108 participants in the micro-ITT NTF-S population (i.e. approximately 81 participants on gepotidacin and 27 on nitrofurantoin). Enrolment will continue until the approximate target number of participants in the micro-ITT NTF-S Population has been reached. This study will be conducted at multiple sites in Japan.

**Note**: Enrolled means a participant's, or their legally acceptable representative's, agreement to participate in a clinical study following completion of the informed consent process. Potential participants who are screened for the purpose of determining eligibility for the study, but do not participate in the study, are not considered enrolled, unless otherwise specified by the protocol. A participant will be considered enrolled if the informed consent is not withdrawn prior to participating in any study activity after screening.

#### 6. SUPPORTING DOCUMENTATION

## 6.1. Appendix 1 Study Population Analyses

Unless otherwise specified, the study population analyses will be based on the ITT and, micro-ITT NTF-S Population. A summary of the number of participants in each of the participant level analysis set will be provided.

#### 6.1.1. Study Population

A summary of the number of participants included in each population will be displayed based on the Screened Population. In addition, a summary and listing of exclusions from study population will be produced based on the ITT population.

## 6.1.2. Participant Disposition

A summary of the number and percentage of participants who completed the study as well as those who prematurely withdrew from the study will be provided. Reasons for study withdrawal will be summarized. Reasons for study withdrawal will be listed.

A summary of study intervention status will be provided. This display will show the number and percentage of participants who have completed the study intervention and the ToC visit or have discontinued the study intervention prematurely, as well as primary reasons for discontinuation of study intervention and the ToC visit.

A summary of the number and percentage of participants who passed screening and entered the study, who failed screening and therefore were not entered into the study, and participants who met eligibility criteria but were not needed will be provided along with the reasons for screen failure. The number of participants will be summarized by Country, Site Id and Investigator Id based on micro-ITT NTF-S Population.

## 6.1.3. Demographic and Baseline Characteristics

The demographic characteristics including age, gender, ethnicity, height/weight, BMI at screening and race will be summarized with descriptive statistics. In addition, the following age categories will be summarized: <18, 18-64 and >=65 based on the ITT and micro-ITT NTF-S populations. The listing of demographic characteristics will be produced as well.

A summary of baseline characteristics will be provided as follows. Data will be listed and summarized using descriptive statistics or frequency counts and percentages as applicable.

| Analysis set | Baseline characteristics |
|---|---|
| ITT Population | Cardiovascular family history |
| ITT, and micro-ITT | Actual randomization strata as per IRT system |
| NTF-S Populations | Age category |
| | Baseline acute cystitis recurrence |
| | Age category as per cCRF (<=50 years, >50 years) |
| | Baseline acute cystitis recurrence |
| | The number of episodes of uncomplicated UTI in the past 3 months, 3-6 months |
| | and 6-12 months. |
| | Baseline renal impairment category (refer to Section 6.2.2.2 for the details) |
| | Baseline quantitative bacterial counts by uropathogen |
| | Number of participants with at least one baseline qualifying uropathogen identified |
| | by uropathogen. |
| | Number of baseline uropathogens identified per participant |
| | Number of baseline qualifying uropathogens identified per participant |
| | Baseline clinical symptom score |
| Micro-ITT Population | Baseline qualifying uropathogens (including phenotypic and genotypic |
| | subcategories) |
| | Baseline qualifying uropathogens by species and group (e.g. Klebsiella spp., other |
| | Enterobacterales, gram-negative nonfermenters, gram-positive species) |
| | The proportion in the above summaries is calculated using the total number of baseline |
| | qualifying uropathogens as denominator. Note that for the participants who have the same |
| | species of more than one baseline qualifying uropathogens (e.g. 2 <i>E coli.</i> ), this will be |
| | counted multiple times. For example, suppose a participant has 2 identical <i>E coli.</i> and |
| | another participant has 1 E coli. and 1 Klebsiella spp. For the proportion of E coli over both |
| | patients is 0.75 (3/4). |

Past medical conditions and current medical conditions as of screening will be summarized respectively based on the ITT Population and micro-ITT NTF-S Population. If the reported medical condition was resolved before screening, this will be regarded as past medical condition. Otherwise, this will be regarded as current medical condition.

Substance use, including smoking history, cigarettes per day, alcohol and caffeine consumption will be summarized based on the ITT Population.

#### 6.1.4. Protocol Deviations

Important protocol deviations will be summarized based on ITT Population.

Protocol deviations will be tracked by the study team throughout the conduct of the study. These protocol deviations will be reviewed to identify those considered as important as follows:

• Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations (where possible without knowing the study intervention details) are captured and categorised in the protocol deviations dataset.

• This dataset will be the basis for the summaries of important protocol deviations.

In addition to the overall summary of important protocol deviations, separate summaries will be produced for important protocol deviations related to COVID-19 based on the ITT Population. Listings of important protocol deviations and subjects with inclusion/exclusions criteria deviations will be produced.

#### 6.1.5. Prior and Concomitant Medications

The analysis is based on the ITT and micro-ITT NTF-S Populations.

Prior and concomitant medications will be coded using WHO Drug dictionaries. The summary of concomitant medications will be provided by Anatomical Therapeutic Chemical (ATC) classification Level 1 and ingredient. Note that multi-ingredient medications will be summarized for a combination of ingredients. Listing of prior and concomitant medications will be produced.

Separate summaries of prior and concomitant medications will be provided for systemic antibiotics as well. An antibiotic is considered systemic if the route is oral, subcutaneous, intramuscular, intravenous, or rectal.

#### 6.1.6. Study Intervention Compliance

Refer to Section 4.6.1.

## 6.1.7. Additional Analyses Due to the COVID-19 Pandemic

A participant is defined as having a suspected, probable or confirmed COVID-19 infection during the study if the answer is "Confirmed", "Probable" or "Suspected" to the case diagnosis question from the COVID-19 coronavirus infection assessment eCRF. Numbers of participants with a suspected, probable or confirmed COVID-19 infection, and of COVID-19 test results will be summarized based on the Safety Population.

Additionally, if greater than 30 participants have a suspected, probable of confirmed COVID-19 infection, the following data displays will be produced:

- Summary of current (and/or past) medical conditions for participants with COVID-19 adverse events.
- Summary of baseline characteristics for participants with COVID-19 adverse events.

## 6.2. Appendix 2 Data Derivations Rule

## 6.2.1. Efficacy

## 6.2.1.1. Microbiological Outcome and Response

Microbiological response by Baseline Qualifying Uropathogen will be derived at Ontherapy, TOC and Follow-up Visits according to Table 7, Table 8 and Table 9. Only start date (not time) of antibiotics use will be considered when deriving the outcome and response.

Participant-level microbiological outcome and response will be derived at On-therapy, TOC and Follow-up Visits according to Table 10.

Microbiological outcome by New Qualifying Uropathogen will be derived at On-therapy Visit according to Table 11, Table 12 and Table 13.

Table 7 Microbiological Outcome by Baseline Qualifying Uropathogen at the On-Therapy Visit

| Defining Criteria | Outcome |
|---|---|
| A quantitative urine culture taken at the On-therapy Visit | Microbiological eradication |
| shows that the qualifying bacterial uropathogen | |
| recovered at Baseline is reduced to <103 CFU/mL, | |
| without the participant receiving other systemic | |
| antimicrobials before the On-therapy Visit | |
| A quantitative urine culture taken at the On-therapy Visit | Microbiological persistence |
| shows that the qualifying bacterial uropathogen | |
| recovered at Baseline grows ≥ 10 <sup>3</sup> CFU/mL, without the | |
| participant receiving other systemic antimicrobials | |
| before the On-therapy Visit | |
| The On-therapy urine culture result is missing, or | Unable to determine |
| The participant received other systemic | |
| antimicrobials before the Ontherapy Visit | |

CFU=colony-forming units.

Table 8 Microbiological Outcome and Response by Baseline Qualifying Uropathogen at the Test of Cure Visit

| Defining Criteria | Outcome | Response |
|---|---|---|
| Participants considered microbiological failures at the TOC Visit will also be considered microbiological failures at | | |
| the Follow-up Visit. | · | |
| A quantitative urine culture taken at the TOC Visit | Microbiological eradication | Microbiological success |
| shows reduction of the qualifying bacterial | | |
| uropathogen recovered at Baseline to <10 <sup>3</sup> CFU/mL, | | |
| without the participant receiving other systemic | | |
| antimicrobials before the TOC Visit | | |
| A quantitative urine culture taken at the TOC Visit | Microbiological persistence | Microbiological failure |
| shows that the qualifying bacterial uropathogen | | |
| recovered at Baseline, and which was also shown to | | |
| persist or unable to determine at the On-therapy Visit, | | |
| grows ≥10³ CFU/mL, without the participant receiving | | |
| other systemic antimicrobials before the TOC Visit | | |

| Defining Criteria | Outcome | Response |
|---|---|---|
| A quantitative urine culture taken at the TOC Visit | Microbiological recurrence | Microbiological failure |
| shows that the qualifying bacterial uropathogen | | |
| recovered at Baseline, and which was also shown to | | |
| be eradicated at the On-therapy Visit, grows ≥103 | | |
| CFU/mL, without the participant receiving other | | |
| systemic antimicrobials before the TOC Visit | | |
| The TOC urine culture result is missing, or | Unable to determine | Microbiological failure |
| The participant received other systemic | | |
| antimicrobials before the TOC Visit | | |

CFU=colony-forming units; TOC=Test-of-Cure.

Table 9 Microbiological Outcome and Response by Baseline Qualifying Uropathogen at the Follow Up Visit

| Defining Criteria | Outcome | Response |
|---|---|---|
| Participants considered microbiological failures at the TOC Visit will also be considered microbiological failures at | | |
| the Follow-up Visit. | T | _ |
| A quantitative urine culture taken at the Follow-up Visit | Sustained microbiological | Microbiological success |
| shows reduction of the qualifying bacterial uropathogen | eradication | |
| recovered at Baseline to <10 <sup>3</sup> CFU/mL, following | | |
| microbiological eradication at the TOC Visit, without the | | |
| participant receiving other systemic antimicrobials before the Follow-up Visit | | |
| A quantitative urine culture taken at the Follow-up Visit | Microbiological recurrence | Microbiological failure |
| shows that the qualifying bacterial uropathogen recovered | Wildiobiological recuirence | Wilciobiological failule |
| at Baseline grows ≥ 10 <sup>3</sup> CFU/mL, following | | |
| microbiological eradication at the TOC Visit, without the | | |
| participant receiving other systemic antimicrobials before | | |
| the Follow-up Visit | | |
| A quantitative urine culture taken at the Follow-up Visit | Microbiological persistence | Microbiological failure |
| shows that the qualifying bacterial uropathogen recovered | | |
| at Baseline grows ≥ 10³ CFU/mL, and also did not | | |
| achieve an outcome of microbiological eradication at the | | |
| TOC Visit, without the participant receiving other systemic | | |
| antimicrobials before the Follow-up Visit | | |
| A quantitative urine culture taken at the Follow-up Visit | Delayed | Microbiological failure |
| shows reduction of the qualifying bacterial uropathogen | microbiological | |
| recovered at Baseline to <10 <sup>3</sup> CFU/mL, and also did not | eradication | |
| achieve an outcome of microbiological eradication at the TOC Visit, without the participant receiving other systemic | | |
| antimicrobials before the Follow-up Visit | | |
| The Follow-up urine culture result is missing, or | Unable to determine | Microbiological failure |
| The participant received other systemic | | Milorobiological fallato |
| antimicrobials before the Follow-up Visit | | |
| antimicrobialo bololo tilo i ollow ap violt | l | |

CFU=colony-forming units; TOC=Test-of-Cure.

Table 10 Participant-Level Microbiological Outcome and Response Definitions per Study Visit

| Defining Criteria at the On-Therapy Visit | Outcome | Response |
|---|---|---|
| All qualifying baseline uropathogens have a microbiological outcome | Microbiological | NA |
| of eradication at On-therapy | eradication | |
| At least one qualifying baseline uropathogen has an outcome of | Microbiological | NA |
| persistence at On-therapy | persistence | |
| All qualifying baseline uropathogen outcomes are unable to | Unable to determine | NA |
| determine at On-therapy | | |
| Defining Criteria at the TOC Visit | Outcome | Response |
| All qualifying baseline uropathogens have a microbiological outcome | Microbiological | Microbiological |
| of eradication at TOC | eradication | success |
| At least one qualifying baseline uropathogen has an outcome of | Microbiological | Microbiological |
| persistence at TOC | persistence | failure |
| At least one qualifying baseline uropathogen has an outcome of | Microbiological | Microbiological |
| recurrence and none have an outcome of persistence at TOC | recurrence | failure |
| All qualifying baseline uropathogen outcomes are unable to | Unable to determine | Microbiological |
| determine at TOC | | failure |
| Defining Criteria at the Follow-up Visit | Outcome | Response |
| All qualifying baseline uropathogens have a microbiological outcome | Sustained | Microbiological |
| of sustained eradication at Follow-up | microbiological | success |
| | eradication | |
| At least one qualifying baseline uropathogen has an outcome of | Microbiological | Microbiological |
| recurrence and none have an outcome of persistence at Follow-up | recurrence | failure |
| At least one qualifying baseline uropathogen has an outcome of | Microbiological | Microbiological |
| persistence at Follow-up | persistence | failure |
| At least one qualifying baseline uropathogen has an outcome of | Delayed microbiological | Microbiological |
| delayed eradication and none have an outcome of persistence or | eradication | failure |
| recurrence at Follow-up | | |
| All qualifying baseline uropathogen outcomes are unable to | Unable to determine | Microbiological |
| determine at Follow-up | | failure |

NA=Not applicable; TOC=Test-of-Cure.

Table 11 Microbiological Outcome by New Qualifying Uropathogen at the On Therapy Visit

| Defining Criteria | Outcome |
|-----------------------------------------------------------|-----------------|
| A new qualifying bacterial uropathogen, not identified at | New uropathogen |
| Baseline, is documented by quantitative urine culture at | |
| the On-therapy Visit | |

# Table 12 Microbiological Outcome by New Qualifying Uropathogen at the Test-of-Cure Visit

| Defining Criteria | Outcome |
|---|---|
| A new qualifying bacterial uropathogen, not identified at Baseline, is documented by quantitative urine culture at the Test-of-Cure Visit in a participant who did not achieve a clinical outcome of clinical resolution at the | New infection |
| Test-of-Cure Visit | |
| A new qualifying bacterial uropathogen, not identified at Baseline, is documented by quantitative urine culture at the Test-of-Cure Visit in a participant who did achieve a clinical outcome of clinical resolution at the Test-of-Cure Visit | Colonization |

Table 13 Microbiological Outcome by New Qualifying Uropathogen at the Follow up Visit

| Defining Criteria | Outcome |
|------------------------------------------------------------|---------------|
| A new qualifying bacterial uropathogen, not identified at | New infection |
| Baseline, is documented by quantitative urine culture at | |
| the Follow-up Visit in a participant who did not achieve a | |
| clinical resolution at the Follow-up Visit | |
| A new qualifying bacterial uropathogen, not identified at | Colonization |
| Baseline, is documented by quantitative urine culture at | |
| the Follow-up Visit in a participant who did achieve a | |
| clinical resolution at the Follow-up Visit | |

## 6.2.1.2. Clinical Outcome and Response

Clinical signs and symptoms of acute cystitis will be recorded based on participant interview per the SoA (Protocol Section 1.3) using the scoring system and instructions (Table 14). The total cumulative symptom score is derived by summing the score for each individual sign and symptom. If any individual sign and symptom scores are missing, then total symptom score will also be missing.

At TOC, success is defined as normal presentation of signs and symptoms with a total cumulative symptom score of zero. Clinical outcome and response will be derived at Ontherapy (Table 15), TOC (Table 16) and Follow-up (Table 17) Visits. Note that "resolution", "improvement" and "worsening or no change" in total symptom score as used in the tables below are defined as:

- "Resolution": Total cumulative symptom score is zero.
- "Improvement": Change from baseline in total cumulative symptom score is less than zero.
- "Worsening or no change": Change from baseline in total cumulative symptom score is greater than or equal to zero.

Note that only start date of antibiotics use will be considered when deriving the outcome and response.

Table 14 Clinical Signs and Symptoms Scoring System

| Clinical Signs and | None | Mild Symptom is easily tolerated, causing minimal discomfort and not interfering with everyday activities | Moderate Symptom is sufficiently discomforting to interfere with normal everyday activities | Severe<br>Symptom prevents<br>normal everyday<br>activities |
|---|---|---|---|---|
| Symptoms | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
| Dysuria | | | | |
| Frequency | | | | |
| Urgency | | | | |
| Lower abdominal or suprapubic pain | | | | |

## Table 15 Clinical Outcome at the On-Therapy Visit

| Defining Criteria | Outcome <sup>a</sup> |
|---|---|
| Resolution of signs and symptoms of acute cystitis | Clinical resolution |
| present at Baseline (and no new signs and symptoms), | |
| without the participant receiving other systemic | |
| antimicrobials not for the current infection before the | |
| On-therapy Visit and also without receiving an other | |
| systemic antimicrobials for the current infection prior to | |
| or at the On-therapy Visit. | |
| Improvement in total symptom scores from Baseline, but | Clinical improvement |
| not complete resolution, without the participant receiving | |
| other systemic antimicrobials (not for the current | |
| infection) before the On-therapy Visit and also without | |
| receiving an other systemic antimicrobials for the current | |
| infection prior to or at the On-therapy Visit. | |
| Worsening or no change in total symptom scores from | Clinical worsening |
| Baseline or the participant received other systemic | |
| antimicrobials for the current infection prior to or on the | |
| date of the On-therapy Visit (if the date of On-therapy | |
| Visit is missing, the end date of the analysis window will | |
| be used as the date of On-therapy visit) | |
| <ul> <li>The Baseline score is missing (unless On-therapy</li> </ul> | Unable to determine |
| score is 0 and no antibiotics use (either not for | |
| current infection or for current infection) then | |
| outcome will be clinical resolution OR unless | |
| Clinical Worsening outcome criteria were met then | |
| outcome will be Clinical worsening), or | |
| <ul> <li>The On-therapy assessment is missing, <u>(unless</u></li> </ul> | |
| clinical worsening outcome criteria were met then | |
| outcome is worsening) or | |
| The participant received other systemic | |
| antimicrobials not for the current infection prior to | |

| Defining Criteria | Outcomea |
|---------------------------------------------------|----------|
| the assessment (unless clinical worsening outcome | |
| criteria were met) | |

a. A study physician or otherwise appropriately medically trained staff will determine the individual clinical signs and symptoms scores for acute cystitis (Table 14), which will then be used to programmatically determine the clinical outcome. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible.

The text with underline is additional clarification to derive the clinical outcome in addition to the protocol table.

Table 16 Clinical Outcome and Response at the Test-of-Cure Visit

| Defining Criteria | Outcomea | Response |
|---|---|---|
| Resolution of signs and symptoms of acute cystitis present at Baseline (and no new signs or symptoms), without the participant receiving other systemic antimicrobials not for the current infection before the TOC Visit and also without receiving an other systemic antimicrobials for the current infection prior to or at the TOC Visit | Clinical resolution | Clinical success |
| Improvement in total symptom scores from Baseline, but not complete resolution, without the participant receiving other systemic antimicrobials not for the current infection before the TOC Visit and also without receiving an other systemic antimicrobials for the current infection prior to or at the TOC Visit | Clinical improvement | Clinical failure |
| Worsening or no change in total symptom scores from Baseline or the participant received other systemic antimicrobials for the current infection before or on the date of the TOC Visit (if the date of TOC Visit is missing, the end date of the analysis window will be used as the date of TOC visit) | Clinical worsening | Clinical failure |
| The Baseline score is missing (unless TOC score is 0 and no antibiotics use (either not for current infection or for current infection) then outcome will be clinical resolution OR unless Clinical worsening outcome criteria were met then outcome will be Clinical worsening), or The TOC assessment is missing (unless clinical worsening outcome criteria were met then outcome is worsening), or The participant received other systemic antimicrobials not for the current infection prior to the assessment (unless clinical worsening criteria were met) | Unable to determine | Clinical failure |

TOC = Test-of-Cure

a. A study physician or otherwise appropriately medically trained staff will determine the individual clinical signs and symptoms scores for acute cystitis (Table 14), which will then be used to programmatically determine the clinical outcome. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible.

The text with underline is additional clarification to derive the clinical outcome and response in addition to the protocol table.

Table 17 Clinical Outcome and Response at the Follow-up Visit

| Defining Criteria | Outcome <sup>a</sup> | Response |
|---|---|---|
| Resolution of signs and symptoms of acute cystitis | Sustained clinical resolution | Clinical success |
| demonstrated at the TOC Visit persist at the | | |
| Follow-up Visit (and no new signs and symptoms), | | |
| without the participant receiving other systemic | | |
| antimicrobials not for the current infection before | | |
| the Follow-up Visit and also without receiving an | | |
| other systemic antimicrobials for the current | | |
| infection prior to or at the Follow Up Visit | | |
| Resolution of signs and symptoms of acute cystitis | Delayed clinical resolution | Clinical failure |
| present at Baseline (and no new signs or | 20.0,000 000 | |
| symptoms), after clinical failure at TOC, without | | |
| the participant receiving other systemic | | |
| antimicrobials not for the current infection before | | |
| the Follow-up Visit and also without receiving an | | |
| other systemic antimicrobials for the current | | |
| infection prior to or at the Follow-Up Visit | | |
| Improvement in total symptom scores from | Clinical improvement | Clinical failure |
| Baseline, but not complete resolution after clinical | Oliffical Improvement | Oliffical failure |
| failure at the TOC visit, without the participant | | |
| receiving other systemic antimicrobials not for the | | |
| current infection before the Follow-up Visit and | | |
| also without receiving an other systemic | | |
| antimicrobials for the current infection prior to or at | | |
| the Follow-Up Visit | | |
| Worsening or no change in total symptom scores | Clinical worsening | Clinical failure |
| at Follow-up compared to Baseline after clinical | Olimical Worserling | Oliffical failure |
| failure at TOC, or the participant received other | | |
| systemic antimicrobials for the current infection | | |
| before or on the date of the Follow-up Visit (if the | | |
| date of Follow-Up Visit is missing, the end date of | | |
| the analysis window will be used as the date of | | |
| Follow-Up visit) | | |
| Signs and symptoms of acute cystitis reoccur at | Clinical recurrence | Clinical failure |
| the Follow-up Visit (can be improved (but not | Official recurrence | Oliffical failure |
| resolution) OR worsening or no change from | | |
| baseline i.e., (1) change from baseline at Follow- | | |
| Up visit < 0 AND score is not 0 at Follow-Up Visit | | |
| (2) change from baseline at the Follow-Up visit >= | | |
| 0) after clinical success at TOC without the | | |
| participant receiving an other systemic | | |
| antimicrobials for the current infection prior to or at | | |
| the Follow-Up visit | | |
| The Baseline score is missing (unless Follow- | Unable to determine | Clinical failure |
| Up score is 0 and no antibiotics use (either | onable to determine | Oliriloar fallaro |
| not for current infection or for current | | |
| infection) then outcome will be clinical | | |
| resolution (delayed or sustained as | | |
| appropriate) OR unless Clinical worsening | | |
| outcome criteria were met then outcome will | | |
| be clinical worsening), or | | |
| The Follow-up assessment is missing (unless) | | |
| clinical worsening outcome criteria were met | | |

| Defining Criteria | Outcome <sup>a</sup> | Response |
|---|---|---|
| The participant received other systemic antimicrobials not for the current infection prior to the assessment (unless the clinical worsening or recurrence outcome criteria were met) | | · |

TOC = Test-of-Cure

a. A study physician or otherwise appropriately medically trained staff will determine the individual clinical signs and symptoms scores for acute cystitis (Table 14), which will then be used to programmatically determine the clinical outcome. The same scorer will be used at all assessment time points for each participant, on all occasions, whenever possible.

The text with underline is additional clarification to derive the clinical outcome in addition to the protocol table.

## 6.2.1.3. Fold change on susceptibility

Fold change will be used to describe how much the MIC for gepotidacin and nitrofurantoin changes between baseline and subsequent visits for the same bacterial species from the same participant based on the broth microdilution results. Fold change will be calculated (in doubling dilutions) as the ratio of the MIC at the subsequent visit to the MIC at Baseline Visit. However, ratio of 1 will be reported as 0-fold ratio. Ratio less than 1 will be reported in reciprocal with negative sign (e.g. ratio of 0.5 will be reported as -2 fold). Examples:

| Baseline MIC (mcg/mL) | Post-baseline MIC (mcg/mL) | Fold-change |
|-----------------------|-------------------------------------|---------------|
| 1 | 1 | 0-fold |
| 1 | 2 | 2-fold |
| 1 | 4 | 4-fold |
| 1 | 8 | 8-fold |
| 1 | 16 | 16-fold |
| 1 | 0.5 | - 2-fold |
| 1 | 0.25 | - 4-fold |
| 1 | >32 | >/=64-fold |
| 1 | >/=32 | >/=32-fold |
| 1 | <0.125 | >/= - 16-fold |
| 1 | =0.125</td <td>&gt;/= - 8-fold</td> | >/= - 8-fold |

#### 6.2.1.4. MIC50 and MIC90

MIC50 and MIC90 are defined as the 50<sup>th</sup> and 90<sup>th</sup> percentile of the MIC values. They will only be reported if the number of uropathogens is larger or equal to 10. MICxx is defined as follows.

$$MICxx = \min_{j} \{x_{j}; \hat{F}(x_{j}) \ge xx\%\}$$
, where  $x_{j}$  is MIC value and  $\hat{F}(\cdot)$  is empirical cumulative distribution.

For an even number of samples, the MIC50 is the next one above the median. Similar algorithm applied to MIC90.

# 6.2.1.5. Investigator-Assessed Clinical Response

| Definitions | Clinical Response |
|---|---|
| Sufficient resolution of acute cystitis signs and symptoms such that no additional systemic | Clinical Success |
| antimicrobial therapy is required for the current infection | |
| Participant met any one of the criteria below: | Clinical Failure |
| No apparent response to treatment (persistence or progression of any pretreatment) | |
| clinical signs and symptoms) | |
| Use of additional systemic antibiotic(s) for the current infection | |
| Death related to acute cystitis prior to the visit | |
| Determination of clinical response could not be made at the visit for any of the following | Indeterminate |
| reasons: | |
| Participant was lost to follow-up and/or the clinical assessment was not undertaken | |
| Use of confounding systemic antibiotic(s) for another infection | |
| Death prior to the visit where acute cystitis was clearly noncontributory | |

Missing data will be handled based on the table below.

| Scenario | Date of data<br>at EW (early<br>withdrawal)<br>Visit | Response at EW visit | Reason for response at EW visit | Start date of<br>Antibiotics<br>use for uUTI | Derivation of data |
|---|---|---|---|---|---|
| Missing at TOC | Date < 17 days<br>+ baseline | Clinical Failure OR Indeterminate | "Death" is contained | NA | Same as data at EW visit |
| Missing at TOC | Any date | Clinical Failure | "Use of additional systemic antibiotic(s) for the current infection" | Baseline <=<br>date <= 17<br>days +<br>baseline | Same as data at EW visit |
| Missing at Follow-Up | Date < 31 days<br>+ baseline | Clinical Failure OR Indeterminate | "Death" is contained | NA | Same as data at EW visit |
| Missing at<br>Follow-Up | Any date | Clinical Failure | "Use of additional systemic antibiotic(s) for the current infection" | Baseline <=<br>date <= 31<br>days +<br>baseline | Same as data at EW visit |
| Any other m | issing other than th | Response: Indeterminate/missing Reason: Participant was lost to follow-up and/or the clinical assessment was not undertaken/missing | | | |



## **6.2.2.** Safety

## **6.2.2.1.** Adverse Events of Special Interest

Cardiovascular (CV) AEs, gastrointestinal (GI) AEs, C. difficile AEs, and AEs related to Acetylcholinesterase Inhibition (AChE-I) as determined by algorithm will be considered AESIs.

## **Clostridium difficile AESIs**

AEs will be regarded as C. difficile AESIs if the preferred terms are either *Clostridium difficile* infection or *Clostridium difficile* colitis.

# **Cardiovascular and Gastrointestinal AESIs**

| Gastrointestinal AESIs are defined as AEs with a "Gastrointestinal disorders" SOC. AEs will be regarded as Cardiovascular AESIs if the preferred terms are any one of the following PTs below. <b>Term</b> | Code | Term | Code |
|---|---|---|---|
| Degenerative aortic valve disease | 10075846 | Tachycardia | 10043071 |
| Supraventricular extrasystoles | 10042602 | Ventricular tachyarrhythmia | 10065341 |
| Rebound tachycardia | 10067207 | Torsade de pointes | 10044066 |
| Cardio-respiratory arrest neonatal | 10007618 | Fascicular block | 10086740 |
| Cardiac flutter | 10052840 | Lown-Ganong-Levine syndrome | 10024984 |
| Paroxysmal arrhythmia | 10050106 | Conduction disorder | 10010276 |
| Cardiac death | 10049993 | Congenital supraventricular tachycardia | 10082343 |
| Atrial conduction time prolongation | 10064191 | Pacemaker generated arrhythmia | 10053486 |
| Neonatal bradyarrhythmia | 10082054 | Wolff-Parkinson-White syndrome | 10048015 |
| Bradycardia foetal | 10006094 | Long QT syndrome | 10024803 |
| Neonatal sinus bradycardia | 10082188 | Parasystole | 10033929 |
| Sinus bradycardia | 10040741 | Cardiac arrest neonatal | 10007516 |
| Marshall-White syndrome | 10088084 | Foetal tachyarrhythmia | 10077575 |
| Junctional ectopic tachycardia | 10074640 | Neonatal sinus tachycardia | 10082191 |
| Ventricular fibrillation | 10047290 | Congenital tricuspid valve stenosis | 10010656 |
| Ventricular parasystole | 10058184 | Parachute mitral valve | 10064192 |
| Pulseless electrical activity | 10058151 | Stroke in evolution | 10059613 |
| Accessory cardiac pathway | 10067618 | Subarachnoid haemorrhage | 10042316 |
| Sinoatrial block | 10040736 | Ischaemic cerebral infarction | 10060840 |
| Paroxysmal atrioventricular block | 10077503 | Spinal subdural haematoma | 10050164 |
| Ogden syndrome | 10082376 | Thrombotic stroke | 10043647 |
| Familial atrial fibrillation | 10088317 | Pituitary infarction | 10035092 |
| Nodal rhythm | 10029470 | Cerebral haemorrhage neonatal | 10008112 |
| Bundle branch block left | 10006580 | Cerebral haemorrhage | 10008111 |
| Precerebral artery embolism | 10085250 | Claude's syndrome | 10085447 |
| Cerebral septic infarct | 10070671 | Vertebrobasilar stroke | 10082484 |
| Cerebellar ischaemia | 10068621 | Intraoperative cerebral artery occlusion | 10056382 |
| Pseudostroke | 10078090 | Cerebral gas embolism | 10070813 |
| Basal ganglia stroke | 10071043 | Brain stem thrombosis | 10062573 |
| Lacunar infarction | 10051078 | Basal ganglia haemorrhage | 10067057 |
| Ruptured cerebral aneurysm | 10039330 | Vertebral artery perforation | 10075735 |
| Malignant middle cerebral artery syndrome | 10086546 | Carotid artery perforation | 10075728 |
| Cerebral artery perforation | 10075734 | Ischaemic stroke | 10061256 |

| Gastrointestinal AESIs are defined as | | | |
|---|---|---|---|
| AEs with a "Gastrointestinal disorders" | | | |
| SOC. AEs will be regarded as | Code | Term | Code |
| Cardiovascular AESIs if the preferred | Code | Term | Code |
| terms are any one of the following PTs | | | |
| below. Term | | | |
| Spinal cord haemorrhage | 10048992 | Cerebral arteriovenous malformation | 10008086 |
| | | haemorrhagic | |
| Subarachnoid haematoma | 10076701 | Cerebrovascular disorder | 10008196 |
| Mitral valve disease | 10061532 | Myxomatous mitral valve degeneration | 10077377 |
| Pulmonary oil microembolism | 10069388 | Mitral valve stenosis | 10027733 |
| Heritable pulmonary arterial hypertension | 10085244 | Pulmonary tumour thrombotic microangiopathy | 10079988 |
| Cor pulmonale acute | 10010969 | Pulmonary venous thrombosis | 10037459 |
| Neonatal pulmonary hypertension | 10088909 | Cement embolism | 10050484 |
| Pulmonary hypertensive crisis | 10068726 | Pulmonary veno-occlusive disease | 10037458 |
| Pulmonary valve incompetence | 10037448 | Newborn persistent pulmonary hypertension | 10053592 |
| Transient aphasia | 10080106 | Pulmonary valve thickening | 10079337 |
| Subclavian steal syndrome | 10042335 | Capsular warning syndrome | 10067744 |
| Tricuspid valve thrombosis | 10088062 | Tricuspid valve incompetence | 10044640 |
| Tricuspid valve disease mixed | 10086096 | Transmyocardial revascularisation | 10059211 |
| Heart valve stenosis | 10061996 | Deep vein thrombosis postoperative | 10066881 |
| Peripheral revascularisation | 10053351 | Carotid revascularisation | 10072559 |
| Respiratory sinus arrhythmia magnitude | 10079115 | Progressive encephalopathy, | 10086607 |
| increased | | hypsarrhythmia and optic atrophy | |
| | | syndrome | |
| Renal artery revascularisation | 10087816 | Unicuspid aortic valve | 10081548 |
| Acute myocardial infarction | 10000891 | Aortic valve atresia | 10066801 |
| Aortic valve disease | 10061589 | Arrhythmia supraventricular | 10003130 |
| Congenital aortic valve incompetence | 10010370 | Reperfusion arrhythmia | 10058156 |
| Supravalvular aortic stenosis | 10042598 | Heart alternation | 10058155 |
| Arrhythmia neonatal | 10003124 | Timothy syndrome | 10079205 |
| Central bradycardia | 10078310 | Foetal heart rate disorder | 10061158 |
| Sinus arrest | 10040738 | Atrial parasystole | 10071666 |
| Cardiac fibrillation | 10061592 | Atrial tachycardia | 10003668 |
| Trifascicular block | 10044644 | Bifascicular block | 10057393 |
| Accelerated idioventricular rhythm | 10049003 | Sudden cardiac death | 10049418 |
| Ventricular tachycardia | 10047302 | Atrioventricular block complete | 10003673 |
| Bundle branch block right | 10006582 | Sinus node dysfunction | 10075889 |
| Bundle branch block bilateral | 10006579 | Sudden death | 10042434 |
| Bezold-Jarisch reflex | 10076999 | Cardio-respiratory arrest | 10007617 |
| Chronotropic incompetence | 10068627 | Neonatal tachyarrhythmia | 10082055 |
| Gastrointestinal AESIs are defined as | | | |
|---|---|---|---|
| AEs with a "Gastrointestinal disorders" | | | |
| SOC. AEs will be regarded as | | | |
| Cardiovascular AESIs if the preferred | Code | Term | Code |
| terms are any one of the following PTs | | | |
| below. <b>Term</b> | | | |
| Baseline foetal heart rate variability | 10074638 | Bradycardia | 10006093 |
| disorder | | | |
| Inherited cardiac conduction disorder | 10070294 | Congenital heart valve incompetence | 10077594 |
| Ventricular flutter | 10047294 | Mitral valve atresia | 10066800 |
| Straddling tricuspid valve | 10083223 | Congenital tricuspid valve incompetence | 10067887 |
| Extraischaemic cerebral haematoma | 10080347 | Congenital heart valve disorder | 10064086 |
| Central nervous system haemorrhage | 10072043 | Congenital tricuspid valve atresia | 10049767 |
| Vertebral artery thrombosis | 10057777 | Cerebral microembolism | 10078311 |
| Vertebral artery occlusion | 10048965 | Carotid aneurysm rupture | 10051328 |
| Pituitary haemorrhage | 10049760 | Cerebral artery occlusion | 10008089 |
| Thalamic infarction | 10064961 | Cerebellar infarction | 10008034 |
| Cerebellar artery occlusion | 10053633 | Cerebral microinfarction | 10083668 |
| Reversible ischaemic neurological deficit | 10050496 | Post stroke depression | 10070606 |
| Cerebral infarction foetal | 10008119 | Precerebral artery thrombosis | 10074717 |
| Brain stem haemorrhage | 10006145 | Brain stem infarction | 10006147 |
| Medullary compression syndrome | 10087065 | Basal ganglia haematoma | 10077031 |
| Lacunar stroke | 10076994 | Mitral valve incompetence | 10027727 |
| Embolic cerebellar infarction | 10084072 | Pulmonary thrombosis | 10037437 |
| Cerebral artery embolism | 10008088 | Pulmonary microemboli | 10037421 |
| Embolism arterial | 10014513 | Hoigne's syndrome | 10059393 |
| Mitral valve calcification | 10050558 | Post procedural pulmonary embolism | 10063909 |
| Systolic anterior motion of mitral valve | 10076976 | Cor pulmonale | 10010968 |
| Pulmonary embolism | 10037377 | Pulmonary arterial hypertension | 10064911 |
| Embolic pneumonia | 10065680 | Pulmonary artery wall hypertrophy | 10063561 |
| Cor pulmonale chronic | 10010970 | Right ventricular hypertension | 10074301 |
| Lambl's excrescences | 10083691 | Tricuspid valve disease | 10061389 |
| Arrhythmia prophylaxis | 10051305 | Cardiac valve rupture | 10068165 |
| ECG signs of myocardial infarction | 10075299 | Heart valve calcification | 10058968 |
| Bicuspid aortic valve | 10004552 | Cardiac valve discolouration | 10079467 |
| Arrhythmia | 10003119 | Cardiac valve vegetation | 10057651 |
| Atrioventricular node dysfunction | 10084085 | Cerebral revascularisation | 10071508 |
| Ventricular pre-excitation | 10049761 | Aortic valve stenosis | 10002918 |
| Supraventricular tachyarrhythmia | 10065342 | Tachyarrhythmia | 10049447 |
| Cardiac arrest | 10007515 | Sinus arrhythmia | 10040739 |
| Atrioventricular node dispersion | 10077893 | Atrioventricular conduction time shortened | 10068180 |
| Holiday heart syndrome | 10083709 | Postural orthostatic tachycardia syndrome | 10063080 |
| Anomalous atrioventricular excitation | 10002611 | Supraventricular tachycardia | 10042604 |

| Gastrointestinal AESIs are defined as AEs with a "Gastrointestinal disorders" SOC. AEs will be regarded as Cardiovascular AESIs if the preferred terms are any one of the following PTs below. <b>Term</b> | Code | Term | Code |
|---|---|---|---|
| Bundle branch block | 10006578 | Sinusoidal foetal heart rate pattern | 10074643 |
| Adams-Stokes syndrome | 10001115 | Bradyarrhythmia | 10049765 |
| Atrioventricular dissociation | 10069571 | Withdrawal arrhythmia | 10047997 |
| Atrial escape rhythm | 10085756 | Tachycardia paroxysmal | 10043079 |
| Atrial flutter | 10003662 | Wandering pacemaker | 10047818 |
| Cardiac failure congestive | 10007559 | Sinus tachycardia | 10040752 |
| Bicuspid pulmonary valve | 10063730 | Arrhythmic storm | 10067339 |
| Weber's syndrome | 10085448 | Ictal bradycardia syndrome | 10088979 |
| Cerebral haemorrhage foetal | 10050157 | Foetal heart rate acceleration abnormality | 10074642 |
| Spinal epidural haematoma | 10050162 | Pacemaker syndrome | 10051994 |
| Basal ganglia infarction | 10069020 | Atrial standstill | 10087237 |
| Cerebellar embolism | 10067167 | Congenital pulmonary valve disorder | 10061075 |
| Spinal subarachnoid haemorrhage | 10073564 | Congenital pulmonary valve atresia | 10052644 |
| Septic cerebral embolism | 10086435 | Congenital mitral valve stenosis | 10010548 |
| Intracranial tumour haemorrhage | 10022775 | Thalamic stroke | 10087626 |
| Post procedural stroke | 10066591 | Basilar artery perforation | 10075736 |
| Embolic cerebral infarction | 10060839 | Brain stem embolism | 10074422 |
| Meningorrhagia | 10052593 | Lateral medullary syndrome | 10024033 |
| Intraventricular haemorrhage neonatal | 10022841 | Occipital lobe stroke | 10089110 |
| Cerebellar haemorrhage | 10008030 | Intracranial haemorrhage neonatal | 10086946 |
| Internal capsule infarction | 10083408 | Pseudo-occlusion of internal carotid artery | 10085779 |
| Pituitary apoplexy | 10056447 | Cerebral vascular occlusion | 10076895 |
| Cerebellar artery thrombosis | 10008023 | Perinatal stroke | 10073945 |
| Brain stem stroke | 10068644 | Cerebral artery thrombosis | 10008092 |
| Mitral valve thickening | 10079336 | Periventricular haemorrhage neonatal | 10076706 |
| Ischaemic mitral regurgitation | 10077864 | Spinal epidural haemorrhage | 10049236 |
| Mitral perforation | 10068138 | Middle cerebral artery stroke | 10027580 |
| Portopulmonary hypertension | 10067281 | Intraventricular haemorrhage | 10022840 |
| Right-to-left cardiac shunt | 10076605 | Haemorrhagic cerebral infarction | 10019005 |
| Congenital pulmonary hypertension | 10050701 | Cerebral infarction | 10008118 |
| Pulmonary valve calcification | 10057464 | Thrombotic cerebral infarction | 10067347 |
| Pulmonary valve disease | 10061541 | Basilar artery thrombosis | 10063093 |
| Pulmonary valve sclerosis | 10057465 | Myocardial infarction | 10028596 |
| Pulmonary valve stenosis | 10037450 | Septic pulmonary embolism | 10083093 |
| Tricuspid valve prolapse | 10066862 | Alveolar capillary dysplasia | 10077023 |
| Prosthetic cardiac valve thrombosis | 10063176 | Coronary sinus dilatation | 10082615 |
| Heart valve incompetence | 10067660 | Pulmonary venous hypertension | 10085364 |

| AEs with a "Gastrointestinal disorders" SOC. AEs will be regarded as Cardiovascular AESIs if the preferred terms are any one of the following PTs below. Term Cardiac valve disease Prosthetic cardiac valve regurgitation Cardiac valve fatty infiltration Deep vein thrombosis Periprocedural myocardial infarction Cerebrovascular pseudoaneurysm Revascularisation procedure 10084087 Aortic valve prolapse 1002388 Aortic annulus rupture 1004943 Aortic valve thickening 1007958 Williams syndrome 10049644 Atrioventricular extrasystoles 1004907 Ectopic atrial rhythm 10088339 Ventricular arrhythmia 10084072 Nodal arrhythmia 10084087 Code Term Code Todo1902 Tocuspid valve sclerosis 1007958 Tricuspid valve sclerosis 1004988 Tricuspid valve thickening 1004988 Coronary revascularisation 1004988 Revascularisation procedure 1005902 Extrasystoles 10075851 Heart block congenital 1001585 Williams syndrome 10049644 Atrioventricular block second degree 1000367 Ventricular extrasystoles 10071710 BRASH syndrome 10084072 Nodal arrhythmia 10029458 Ventricular arrhythmia 1004728 | Gastrointestinal AESIs are defined as | | | |
|---|---|---|---|---|
| SOC. AEs will be regarded as Cardiovascular AESIs if the preferred terms are any one of the following PTs below. Term Cardiac valve disease Prosthetic cardiac valve regurgitation Cardiac valve fatty infiltration Deep vein thrombosis Periprocedural myocardial infarction Cerebrovascular pseudoaneurysm Revascularisation procedure Aortic valve prolapse Aortic valve prolapse Aortic valve thickening 1007938 Aortic valve prolapse 10061406 Amaurosis fugax 10001903 Tricuspid valve sclerosis 1005746 Cardiac valve thickening 1007933 Tricuspid valve thickening 1007958 Periprocedural myocardial infarction 10079319 Silent myocardial infarction 1004968 Revascularisation procedure 10084091 Foetal cerebrovascular disorder 1005360 Angina unstable 10002388 Aortic annulus rupture 10079581 Aortic valve prolapse 10057454 Subvalvular aortic stenosis 1004243 Aortic valve thickening 10075851 Heart block congenital 1001926 Aortic valve sclerosis 10002917 Extrasystoles 1001585 Williams syndrome 10049644 Atrioventricular block second degree 1000367 Ventricular extrasystoles 10047289 Brugada syndrome 10049029 congenital Lenegre's disease 10071710 BRASH syndrome 10084072 Nodal arrhythmia 1004728 | | | | |
| Cardiovascular AESIs if the preferred terms are any one of the following PTs below. Term Cardiac valve disease 10061406 Amaurosis fugax 1000190: Prosthetic cardiac valve regurgitation 10087802 Tricuspid valve sclerosis 1005746 Cardiac valve fatty infiltration 10087637 Tricuspid valve thickening 1007933: Deep vein thrombosis 10051055 Cardiac valve thickening 1007958: Periprocedural myocardial infarction 10079319 Silent myocardial infarction 1004976: Cerebrovascular pseudoaneurysm 10084087 Coronary revascularisation 1004988: Revascularisation procedure 10084091 Foetal cerebrovascular disorder 1007958: Aortic valve prolapse 10057454 Subvalvular aortic stenosis 1004243 Aortic valve thickening 10075851 Heart block congenital 1001926: Aortic valve sclerosis 10049644 Atrioventricular block second degree 1000367: Ventricular extrasystoles 10047289 Brugada syndrome 1004909 Ectopic atrial rhythm 10088339 Wolff-Parkinson-White syndrome 1004909 Lenegre's disease 10071710 BRASH syndrome 1004728 Ventricular arrhythmia 1004728 | | | | |
| terms are any one of the following PTs below. Term Cardiac valve disease 10061406 Amaurosis fugax 1000190. Prosthetic cardiac valve regurgitation 10087802 Tricuspid valve sclerosis 1005746 Cardiac valve fatty infiltration 10087637 Tricuspid valve thickening 1007933. Deep vein thrombosis 10051055 Cardiac valve thickening 1007958. Periprocedural myocardial infarction 10079319 Silent myocardial infarction 1004976. Cerebrovascular pseudoaneurysm 10084087 Coronary revascularisation 1004988. Revascularisation procedure 10084091 Foetal cerebrovascular disorder 1005360. Angina unstable 10002388 Aortic annulus rupture 1007958. Aortic valve prolapse 10057454 Subvalvular aortic stenosis 1004243. Aortic valve thickening 10075851 Heart block congenital 1001926. Aortic valve sclerosis 10002917 Extrasystoles 1001585. Williams syndrome 10049644 Atrioventricular block second degree 1000367. Ventricular extrasystoles 10047289 Brugada syndrome 1005902. Ectopic atrial rhythm 10088339 Wolff-Parkinson-White syndrome 1004929. Lenegre's disease 10071710 BRASH syndrome 10084072. Nodal arrhythmia 10029458 Ventricular arrhythmia 1004728 | _ | Code | Term | Code |
| below. TermCardiac valve disease10061406Amaurosis fugax10001903Prosthetic cardiac valve regurgitation10087802Tricuspid valve sclerosis1005746Cardiac valve fatty infiltration10087637Tricuspid valve thickening1007933Deep vein thrombosis10051055Cardiac valve thickening1007958Periprocedural myocardial infarction10079319Silent myocardial infarction1004976Cerebrovascular pseudoaneurysm10084087Coronary revascularisation1004988Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture1007958Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital1001926Aortic valve sclerosis10002917Extrasystoles1001585Williams syndrome10049644Atrioventricular block second degree1000367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929Lenegre's disease10071710BRASH syndrome1008407Nodal arrhythmia10029458Ventricular arrhythmia1004728 | · | | | |
| Cardiac valve disease10061406Amaurosis fugax1000190Prosthetic cardiac valve regurgitation10087802Tricuspid valve sclerosis1005746Cardiac valve fatty infiltration10087637Tricuspid valve thickening1007933Deep vein thrombosis10051055Cardiac valve thickening1007958Periprocedural myocardial infarction10079319Silent myocardial infarction1004976Cerebrovascular pseudoaneurysm10084087Coronary revascularisation1004988Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture1007958Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital1001926Aortic valve sclerosis10002917Extrasystoles1001585Williams syndrome10049644Atrioventricular block second degree100367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929Lenegre's disease10071710BRASH syndrome1008407Nodal arrhythmia10029458Ventricular arrhythmia1004728 | , | | | |
| Prosthetic cardiac valve regurgitation10087802Tricuspid valve sclerosis1005746Cardiac valve fatty infiltration10087637Tricuspid valve thickening1007933Deep vein thrombosis10051055Cardiac valve thickening1007958Periprocedural myocardial infarction10079319Silent myocardial infarction1004976Cerebrovascular pseudoaneurysm10084087Coronary revascularisation1004988Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture1007958Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital1001926Aortic valve sclerosis10002917Extrasystoles1001585Williams syndrome10049644Atrioventricular block second degree100367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929Lenegre's disease10071710BRASH syndrome1008407Nodal arrhythmia10029458Ventricular arrhythmia1004728 | | 10061406 | Amaurosis fugax | 10001903 |
| Cardiac valve fatty infiltration10087637Tricuspid valve thickening10079333Deep vein thrombosis10051055Cardiac valve thickening1007958Periprocedural myocardial infarction10079319Silent myocardial infarction1004976Cerebrovascular pseudoaneurysm10084087Coronary revascularisation1004988Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture1007958Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital1001926Aortic valve sclerosis10002917Extrasystoles1001585Williams syndrome10049644Atrioventricular block second degree100367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929congenitalLenegre's disease10071710BRASH syndrome1008407Nodal arrhythmia10029458Ventricular arrhythmia1004728 | | | | |
| Deep vein thrombosis10051055Cardiac valve thickening1007958Periprocedural myocardial infarction10079319Silent myocardial infarction1004976Cerebrovascular pseudoaneurysm10084087Coronary revascularisation1004988Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture1007958Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital1001926Aortic valve sclerosis10002917Extrasystoles1001585Williams syndrome10049644Atrioventricular block second degree1000367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929congenitalLenegre's disease10071710BRASH syndrome1008407Nodal arrhythmia10029458Ventricular arrhythmia1004728 | | | ' | |
| Periprocedural myocardial infarction10079319Silent myocardial infarction1004976Cerebrovascular pseudoaneurysm10084087Coronary revascularisation1004988Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture1007958Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital1001926Aortic valve sclerosis10002917Extrasystoles1001585Williams syndrome10049644Atrioventricular block second degree1000367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929congenitalLenegre's disease10071710BRASH syndrome1008407Nodal arrhythmia10029458Ventricular arrhythmia1004728 | • | | | |
| Cerebrovascular pseudoaneurysm10084087Coronary revascularisation1004988Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture1007958Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital1001926Aortic valve sclerosis10002917Extrasystoles1001585Williams syndrome10049644Atrioventricular block second degree1000367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929congenitalLenegre's disease10071710BRASH syndrome10084073Nodal arrhythmia10029458Ventricular arrhythmia1004728 | • | | _ | |
| Revascularisation procedure10084091Foetal cerebrovascular disorder1005360Angina unstable10002388Aortic annulus rupture10079581Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital10019263Aortic valve sclerosis10002917Extrasystoles10015856Williams syndrome10049644Atrioventricular block second degree1000367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929congenitalcongenitalLenegre's disease10071710BRASH syndrome10084073Nodal arrhythmia10029458Ventricular arrhythmia1004728 | • | | • | |
| Angina unstable10002388Aortic annulus rupture10079586Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital10019263Aortic valve sclerosis10002917Extrasystoles10015856Williams syndrome10049644Atrioventricular block second degree10003677Ventricular extrasystoles10047289Brugada syndrome10059027Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome10049296congenitalcongenital10084077Nodal arrhythmia10029458Ventricular arrhythmia10047286 | , , | | | |
| Aortic valve prolapse10057454Subvalvular aortic stenosis1004243Aortic valve thickening10075851Heart block congenital10019263Aortic valve sclerosis10002917Extrasystoles10015856Williams syndrome10049644Atrioventricular block second degree1000367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929congenitalcongenitalLenegre's disease10071710BRASH syndrome10084073Nodal arrhythmia10029458Ventricular arrhythmia1004728 | | | | |
| Aortic valve thickening 10075851 Heart block congenital 1001926 Aortic valve sclerosis 10002917 Extrasystoles 10015856 Williams syndrome 10049644 Atrioventricular block second degree 1000367 Ventricular extrasystoles 10047289 Brugada syndrome 1005902 Ectopic atrial rhythm 10088339 Wolff-Parkinson-White syndrome 1004929 congenital Lenegre's disease 10071710 BRASH syndrome 10084073 Nodal arrhythmia 10029458 Ventricular arrhythmia 1004728 | | | i i | |
| Aortic valve sclerosis 10002917 Extrasystoles 10015856 Williams syndrome 10049644 Atrioventricular block second degree 1000367 Ventricular extrasystoles 10047289 Brugada syndrome 1005902 Ectopic atrial rhythm 10088339 Wolff-Parkinson-White syndrome 1004929 congenital Lenegre's disease 10071710 BRASH syndrome 10084073 Nodal arrhythmia 10029458 Ventricular arrhythmia 1004728 | • | | | |
| Williams syndrome10049644Atrioventricular block second degree1000367Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome1004929congenitalcongenitalLenegre's disease10071710BRASH syndrome10084073Nodal arrhythmia10029458Ventricular arrhythmia1004728 | | | | |
| Ventricular extrasystoles10047289Brugada syndrome1005902Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome<br>congenital1004929Lenegre's disease10071710BRASH syndrome10084073Nodal arrhythmia10029458Ventricular arrhythmia1004728 | | | | |
| Ectopic atrial rhythm10088339Wolff-Parkinson-White syndrome<br>congenital1004929Lenegre's disease10071710BRASH syndrome10084073Nodal arrhythmia10029458Ventricular arrhythmia1004728 | | | | |
| Lenegre's disease 10071710 BRASH syndrome 10084073 Nodal arrhythmia 10029458 Ventricular arrhythmia 1004728 | | | | |
| Lenegre's disease10071710BRASH syndrome10084073Nodal arrhythmia10029458Ventricular arrhythmia1004728 | Letopic atrial mytim | 10000000 | • | 10043231 |
| Nodal arrhythmia 10029458 Ventricular arrhythmia 1004728 | Lenegre's disease | 10071710 | | 10084073 |
| LEDETAL CARDIAC ARTEST LETIONAL/AND LEARNY REPORTS FOR THE LETION SYNDROME LETIONAL | Foetal cardiac arrest | 10084280 | Early repolarisation syndrome | 10047231 |
| | | | | 10074636 |
| | • | | | 10077926 |
| | | | | 10057526 |
| | | | | 10086078 |
| syndrome | Volumedial develore | 10011201 | | 10000070 |
| | Defect conduction intraventricular | 10012118 | | 10082089 |
| | | | · · | 10056471 |
| | • | | | 10066802 |
| | | | ' | 10037451 |
| | • | | | 10014075 |
| | | | • | 10048964 |
| | | | | 10061038 |
| | , , | | | 10058571 |
| | • | | i ' | 10056237 |
| | • | | | 10053942 |
| | | | | 10018985 |
| | • | | | 10014498 |
| | _ | | | 10089109 |
| | | | | 10076051 |

| Gastrointestinal AESIs are defined as AEs with a "Gastrointestinal disorders" SOC. AEs will be regarded as Cardiovascular AESIs if the preferred terms are any one of the following PTs below. <b>Term</b> | Code | Term | Code |
|---|---|---|---|
| Basilar artery occlusion | 10048963 | Haemorrhagic transformation stroke | 10055677 |
| Cerebellar stroke | 10079062 | Precerebral artery occlusion | 10036511 |
| Inner ear infarction | 10070754 | Brain stem ischaemia | 10006148 |
| Cerebral ischaemia | 10008120 | Cerebral aneurysm perforation | 10075394 |
| Benedikt's syndrome | 10085451 | Thalamus haemorrhage | 10058939 |
| Intracranial haematoma | 10059491 | Carotid arterial embolus | 10007684 |
| Haemorrhagic stroke | 10019016 | Subdural haemorrhage neonatal | 10042365 |
| Cerebral thrombosis | 10008132 | Subarachnoid haemorrhage neonatal | 10042317 |
| Mitral valve disease mixed | 10027724 | Haemorrhagic cerebellar infarction | 10085944 |
| Degenerative mitral valve disease | 10075847 | Cerebrovascular accident | 10008190 |
| Metastatic pulmonary embolism | 10069909 | Mitral valve sclerosis | 10051538 |
| Carcinoid heart disease | 10069010 | Mitral face | 10073380 |
| Cardiac valve replacement complication | 10053748 | Mitral valve prolapse | 10027730 |
| Degenerative multivalvular disease | 10081779 | Obstetrical pulmonary embolism | 10029925 |
| Cardiac valve sclerosis | 10061082 | Anaphylactoid syndrome of pregnancy | 10067010 |
| Cardiac valve abscess | 10064267 | Pulmonary artery thrombosis | 10037340 |
| Respiratory sinus arrhythmia magnitude | 10079114 | Pulmonary hypertension | 10037400 |
| Respiratory sinus arrhythmia magnitude abnormal | 10079117 | Transient ischaemic attack | 10044390 |
| Congenital aortic valve stenosis | 10010371 | Tricuspid valve stenosis | 10044642 |
| Aortic valve calcification | 10050559 | Degenerative tricuspid valve disease | 10078909 |
| Aortic valve incompetence | 10002915 | Tricuspid valve calcification | 10057466 |
| Heyde's syndrome | 10049251 | Post procedural myocardial infarction | 10066592 |
| Aortic valve disease mixed | 10002912 | Respiratory sinus arrhythmia magnitude decreased | 10079116 |
| - | - | Arterial revascularisation | 10084482 |

# **Acetylcholinesterase Inhibition AESIs**

AEs will be regarded as Acetylcholinesterase Inhibition AESIs if the preferred terms are any one of the following PTs below.

| Term | Code | Term | Code |
|---|---|---|---|
| Atrioventricular block first degree | 10003674 | Convulsions local | 10010920 |
| Atonic seizures | 10003628 | Diarrhoea | 10012735 |
| Bradycardia foetal | 10006094 | Status epilepticus | 10041962 |
| Diarrhoea haemorrhagic | 10012741 | Laryngeal dyspnoea | 10052390 |
| Dysarthria | 10013887 | Prophylaxis against bronchospasm | 10054927 |

| Term | Code | Term | Code |
|---|---|---|---|
| Dyspnoea paroxysmal nocturnal | 10013974 | Post procedural diarrhoea | 10057585 |
| Retching | 10038776 | Procedural vomiting | 10066963 |
| Simple partial seizures | 10040703 | Idiopathic generalised epilepsy | 10071081 |
| Sinus bradycardia | 10040741 | Bradycardia | 10006093 |
| Vomiting projectile | 10047708 | Convulsive threshold lowered | 10010927 |
| Self-induced vomiting | 10048636 | Diarrhoea infectious neonatal | 10012744 |
| Hypoglycaemic seizure | 10048803 | Dyspnoea at rest | 10013969 |
| Lennox-Gastaut syndrome | 10048816 | Frequent bowel movements | 10017367 |
| Nocturnal dyspnoea | 10049235 | Haematemesis | 10018830 |
| Atypical benign partial epilepsy | 10056699 | Nausea | 10028813 |
| Hyponatraemic seizure | 10073183 | Tonic convulsion | 10043994 |
| Infantile vomiting | 10075315 | Frontal lobe epilepsy | 10049424 |
| Neonatal sinus bradycardia | 10082188 | Tonic clonic movements | 10051171 |
| Abdominal discomfort | 10000059 | Clonic convulsion | 10053398 |
| Defaecation urgency | 10012110 | Lafora's myoclonic epilepsy | 10054030 |
| Drooling | 10013642 | Psychogenic seizure | 10058895 |
| Epilepsy | 10015037 | Partial seizures | 10061334 |
| Flatulence | 10016766 | Seizure like phenomena | 10071048 |
| Heart rate decreased | 10019301 | Change in seizure presentation | 10075606 |
| Hyperkinesia | 10020651 | Idiopathic partial epilepsy | 10076552 |
| Petit mal epilepsy | 10034759 | Post stroke seizure | 10076981 |
| Psychomotor hyperactivity | 10037211 | Abdominal pain lower | 10000084 |
| Vomiting | 10047700 | Cold sweat | 10009866 |
| Myoclonic epilepsy | 10054859 | Diarrhoea infectious | 10012742 |
| Partial seizures with secondary | 10056209 | Dyspnoea exertional | 10013971 |
| generalisation | | | |
| Alcoholic seizure | 10056347 | Febrile convulsion | 10016284 |
| Therapeutic emesis | 10058324 | Generalised tonic-clonic seizure | 10018100 |
| Faecal vomiting | 10064670 | Night sweats | 10029410 |
| Psychogenic pseudosyncope | 10075190 | Presyncope | 10036653 |
| Central bradycardia | 10078310 | Sweat gland disorder | 10042653 |
| Gastrointestinal disorder | 10017944 | Bradyarrhythmia | 10049765 |
| Hyperemesis gravidarum | 10020614 | Convulsion in childhood | 10052391 |
| Lacrimation decreased | 10023642 | Prophylaxis of nausea and vomiting | 10054133 |
| Vomiting psychogenic | 10047709 | Increased bronchial secretion | 10062530 |
| Wheezing | 10047924 | Transfusion-associated dyspnoea | 10072266 |
| Viral diarrhoea | 10051511 | Hypocalcaemic seizure | 10072456 |
| Epigastric discomfort | 10053155 | Abdominal pain | 10000081 |
| Antidiarrhoeal supportive care | 10055660 | Abdominal pain upper | 10000087 |
| Bronchial hyperreactivity | 10066091 | Bronchospasm | 10006482 |
| Gastrointestinal tract irritation | 10070840 | Gastrointestinal pain | 10017999 |

| Term | Code | Term | Code |
|---|---|---|---|
| Focal dyscognitive seizures | 10079424 | Hyperhidrosis | 10020642 |
| Febrile infection-related epilepsy | 10079438 | Salivary hypersecretion | 10039424 |
| syndrome | | | |
| Neonatal epileptic seizure | 10082068 | Seizure | 10039906 |
| Gelastic seizure | 10082918 | Sweating fever | 10042666 |
| Abdominal tenderness | 10000097 | Syncope | 10042772 |
| Drug withdrawal convulsions | 10013752 | Bradycardia neonatal | 10056471 |
| Dyspnoea | 10013968 | Acetonaemic vomiting | 10058938 |
| Lacrimation increased | 10023644 | Abdominal symptom | 10060926 |
| Seizure anoxic | 10039907 | Cyclic vomiting syndrome | 10062937 |
| Autonomic seizure | 10049612 | Prophylaxis against diarrhoea | 10064065 |
| Benign familial neonatal convulsions | 10067866 | Post-tussive vomiting | 10066220 |
| Hyperglycaemic seizure | 10071394 | Procedural nausea | 10066962 |
| Unilateral bronchospasm | 10072338 | Seizure cluster | 10071350 |
| Faeces soft | 10074859 | Migraine-triggered seizure | 10076676 |
| Irregular breathing | 10076213 | Acute encephalitis with refractory, | 10076948 |
| | | repetitive partial seizures | |
| Asthma | 10003553 | Discoloured vomit | 10079120 |
| Bacterial diarrhoea | 10004016 | Epilepsy with myoclonic-atonic seizures | 10081179 |
| Bronchospasm paradoxical | 10006486 | Seizure prophylaxis | 10081601 |
| - | - | Neonatal seizure | 10082067 |

## 6.2.2.2. Renal impairment

The severity of renal impairment will be evaluated using estimated by creatinine clearance (Ccr).

Severity of renal impairment will be categorized based on creatinine clearance as below (rounded to the nearest integer):

- Normal ( $\geq 90 \, mL/min$ )
- Mild ( $\geq$  60 to 89 mL/min)
- Moderate ( $\geq 30 \text{ to } 59 \text{ mL/min}$ )
- Severe (< 30 *mL/min*)

# **6.2.3.** Criteria for Potential Clinical Importance

# 6.2.3.1. ECG

| ECG Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | N/A | >450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |

# 6.2.3.2. Vital Signs

| Vital Sign Parameter | Units | Potentially Clinically Important Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Pulse Rate | bpm | < 40 | > 110 |

## 6.2.4. Division of Microbiology and Infectious Diseases Adult Toxicity Tables for Adverse Event Assessment

### 6.2.4.1. Laboratory Values

For grading, only numerical criteria will be used in the derivation rules as follows.

### **Adults:**

For adults, laboratory abnormalities will be graded according to the modified US National institute of Allergy and Infectious Diseases Division of Microbiology and Infectious Diseases (DMID) criteria, which is aligned with the global studies (204989 and 212390). Laboratory results are converted to SI units.

| HEMATOLOGY | HEMATOLOGY | | | | | |
|---|---|---|---|---|---|---|
| | Laboratory parameter | Display label | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | Hemoglobin | Hemoglobin (Low) | 9.5 to 10.5 g/dL | 8.0 to 9.4 g/dL | 6.5 to 7.9 g/dL | <6.5 g/dL |
| Absolute Neutrophil Count | Neutrophils | Neutrophils (Low) | 1000 to 1500 /mm <sup>3</sup> | 750 to 999 /mm <sup>3</sup> | 500 to 749 /mm <sup>3</sup> | <500 /mm <sup>3</sup> |
| Platelets | Platelets | Platelets (Low) | 75,000 to 99,999 /mm <sup>3</sup> | 50,000 to 74,999 /mm <sup>3</sup> | 20,000 to 49,999 /mm <sup>3</sup> | <20,000 /mm <sup>3</sup> |
| White Blood Cells | Leukocytes | Leukocytes<br>(High) | 11,000 to 13,000 /mm <sup>3</sup> | 13,001 to 15,000 /mm <sup>3</sup> | 15,001 to 30,000 /mm <sup>3</sup> | >30,000 or <1000 /mm <sup>3</sup> |
| % Polymorphonuclear Leukocytes<br>+ Band Cells | NA | NA | >80% | 90 to 95% | >95% | N/A |
| Abnormal Fibrinogen | NA | NA | Low: 100 to 200 mg/dL<br>High: 400 to<br>600 mg/dL | Low: <100 mg/dL<br>High: >600 mg/dL | Low: <50 mg/dL<br>High: N/A | Fibrinogen associated with gross bleeding or with disseminated coagulation |
| Fibrin Split Product | NA | NA | 20 to 40 mcg/mL | 41 to 50 mcg/mL | 51 to 60 mcg/dL | >60 mcg/dL |
| Prothrombin Time (PT) | NA | NA | 1.01 to 1.25 × ULN | 1.26 to 1.5 × ULN | 1.51 to 3.0 × ULN | >3 × ULN |
| Activated Partial Thromboplastin (APTT) | NA | NA | 1.01 to 1.66 × ULN | 1.67 to 2.33 × ULN | 2.34 to 3 × ULN | >3 ×ULN |
| Methemoglobin | NA | NA | 5.0 to 9.9% | 10.0 to 14.9% | 15.0 to 19.9% | >20% |

N/A=not applicable; ULN=upper limit of normal.

| CHEMISTRIES | CHEMISTRIES | | | | | |
|---|---|---|---|---|---|---|
| | Laboratory parameter | Display label | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | Sodium | Sodium (Low) | 130 to 135 mEq/L | 123 to<br>129 mEq/L | 116 to 122 mEq/L | <116 mEq/L or abnormal sodium with mental status changes or seizures |
| Hypernatremia | Sodium | Sodium (High) | 146 to 150 mEq/L | 151 to<br>157 mEq/L | 158 to 165 mEq/L | >165 mEq/L or abnormal sodium with mental status changes or seizures |
| Hypokalemia | Potassium | Potassium (Low) | 3.0 to 3.4 mEq/L | 2.5 to 2.9 mEq/L | 2.0 to 2.4 mEq/L or intensive replacement therapy of hospitalization required | <2.0 mEq/L or abnormal potassium with paresis, ileus, or life-threatening arrhythmia |
| Hyperkalemia | Potassium | Potassium (High) | 5.6 to 6.0 mEq/L | 6.1 to 6.5 mEq/L | 6.6 to 7.0 mEq/L | >7.0 mEq/L or abnormal potassium with life-threatening arrhythmia |
| Hypoglycemia | Glucose | Glucose (Low) | 55 to 64 mg/dL | 40 to 54 mg/dL | 30 to 39 mg/dL | <30 mg/dL or abnormal glucose with mental status changes or coma |
| Hyperglycemia<br>(nonfasting and no prior<br>diabetes) | Glucose | Glucose (High) | 116 to 160 mg/dL | 161 to<br>250 mg/dL | 251 to 500 mg/dL | >500 mg/dL or abnormal glucose with ketoacidosis or seizures |
| Hypocalcemia (corrected for albumin) | Calcium | Calcium (Low) | 8.4 to 7.8 mg/dL | 7.7 to 7.0 mg/dL | 6.9 to 6.1 mg/dL | <6.1 mg/dL or abnormal calcium with life-threatening arrhythmia or tetany |
| Hypercalcemia (corrected for albumin) | Calcium | Calcium (High) | 10.6 to 11.5 mg/dL | 11.6 to<br>12.5 mg/dL | 12.6 to 13.5 mg/dL | >13.5 mg/dL or abnormal calcium with life-threatening arrhythmia |
| Hypomagnesemia | Magnesium | Magnesium (Low) | 1.4 to 1.2 mEq/L | 1.1 to 0.9 mEq/L | 0.8 to 0.6 mEq/L | <0.6 mEq/L or abnormal magnesium with life-threatening arrhythmia |
| Hypophosphatemia | Phosphate | Phosphate (Low) | 2.0 to 2.4 mg/dL | 1.5 to 1.9 mg/dL<br>or replacement<br>Rx required | 1.0 to 1.4 mg/dL<br>intensive therapy or<br>hospitalization required | <1.0 mg/dL or abnormal phosphate with life-threatening arrhythmia |

| CHEMISTRIES | CHEMISTRIES | | | | | |
|---|---|---|---|---|---|---|
| | Laboratory parameter | Display label | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyperbilirubinemia (when accompanied by any increase in other liver function test) | Bilirubin (when any of AST, ALT and ALP is greater than the upper limit of normal range at the same analysis visit) | Bilirubin (High) | 1.1 to<br><1.25 × ULN | 1.25 to<br><1.5 × ULN | 1.5 to 1.75 × ULN | >1.75 × ULN |
| Hyperbilirubinemia (when other liver function tests are in the normal range) | Bilirubin (when all of AST, ALT and ALP are within the normal range at the same analysis visit) | Bilirubin (High) | 1.1 to <1.5 × ULN | 1.5 to<br><2.0 × ULN | 2.0 to 3.0 × ULN | >3.0 × ULN |
| Blood urea nitrogen | Urea | Urea Nitrogen<br>(High) | 1.25 to 2.5 × ULN | 2.6 to 5 × ULN | 5.1 to 10 × ULN | >10 × ULN |
| Hyperuricemia (uric acid) | NA | NA | 7.5 to 10.0 mg/dL | 10.1 to<br>12.0 mg/dL | 12.1 to 15.0 mg/dL | >15.0 mg/dL |
| Creatinine | Creatinine | Creatinine (High) | 1.1 to 1.5 × ULN | 1.6 to 3.0 × ULN | 3.1 to 6.0 × ULN | >6 × ULN or dialysis required |

Rx=therapy; ULN=upper limit of normal

| ENZYMES | ENZYMES | | | | | |
|---|---|---|---|---|---|---|
| | Laboratory parameter | Display label | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Aspartate<br>aminotransferase<br>(AST) | Aspartate aminotransferase | Aspartate aminotransferase (High) | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alanine<br>aminotransferase<br>(ALT) | Alanine<br>aminotransferase | Alanine aminotransferase (High) | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Gamma to glutamyl transferase (GGT) | NA | NA | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Alkaline<br>Phosphatase | Alkaline<br>Phosphatase | Alkaline Phosphatase (High) | 1.1 to <2.0 × ULN | 2.0 to <3.0 × ULN | 3.0 to 8.0 × ULN | >8.0 × ULN |
| Amylase | NA | NA | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |
| Lipase | NA | NA | 1.1 to 1.5 × ULN | 1.6 to 2.0 × ULN | 2.1 to 5.0 × ULN | >5.1 × ULN |

ULN=upper limit of normal.

| URINALYSIS | | | | | | |
|---|---|---|---|---|---|---|
| | Laboratory parameter | Display label | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Proteinuria | NA | NA | 1+ or<br>200 mg to 1 gm loss/day | 2 to 3+ or<br>1 to 2 gm<br>loss/day | 4+ or<br>2 to 3.5 gm loss/day | Nephrotic syndrome or >3.5 gm loss/day |
| Hematuria | NA | NA | Microscopic only<br><10 RBC/hpf | Gross, no clots >10 RBC/hpf | Gross, with or without clots, or red blood cells casts | Obstructive or required transfusion |

HPF=high powered field; RBC=red blood cells.

### **Adolescent Participants:**

For adolescent participants over 12 years of age and less than 18 years of age, the adult DMID will be applied for all parameters with the exception of serum creatinine which will be graded programmatically according to the modified DMID pediatric toxicity criteria, which is aligned with the global studies (204989 and 212390). Laboratory results are converted to SI units.

| CHEMISTRIES | | | | | | |
|---|---|---|---|---|---|---|
| | Laboratory parameter | Display label | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Creatinine | Creatinine | Creatinine (High) | 1.0 to 1.7 x ULN | 1.8 to 2.4 x ULN | 2.5 to 3.5 x ULN | >3.5 x ULN |

ULN=upper limit of normal.

### 6.2.5. Study Period

Assessments and events will be classified according to the time of occurrence relative to the study intervention period.

**Pre-Intervention** is defined as time prior to the first dose of study intervention.

**On-Intervention** is defined as time from first dose to last date. If time of assessment or study intervention is not collected, the following assessment on the first dose date will be assumed to be taken prior to the first dose and therefore considered pre-intervention: ECG, Lab, and vital signs, and first dose date is considered on-intervention for AE and concomitant medication.

**Post-Intervention** is defined as any time post on-intervention window, i.e. > last dose date.

#### 6.2.5.1. Study Phases for Concomitant medication

| Study Phase | Definition |
|---|---|
| Prior | If medication started prior to the first dose date (or randomized date if first dose date is missing) |
| Concomitant | If medication ended after the first dose date or is ongoing regardless of the start date (or randomized date if first dose date is missing) |

Study phases for concomitant medication will be derived after handling of missing and partial dates for medication (see Section 6.2.9). If a single medication taken on the same date as the first dose date, time will be used to determine if it's prior or concomitant. If time is missing, it will be considered concomitant.

#### 6.2.5.2. Treatment Emergent Flag for Adverse Events

Adverse events are defined as treatment emergent AEs if AE onset date/time is on or after treatment start date/time. That is, study treatment start date/time <= AE start date/time. If time is missing, only date will be compared.

#### 6.2.5.3. Participant and Study Completion

A participant is considered to have completed study treatment if she has taken all doses of the randomly assigned study treatment and also completed the ToC visit. A participant is considered to have completed the study if she has completed all study visits including the Follow-up Visit.

### 6.2.6. Study Day and Reference Dates

The safety reference date is the study intervention start date (or randomization date if not dosed) and will be used to calculate study day for safety measures.

The efficacy reference date is the study intervention start date (or randomization date if not dosed) and will be used to calculate study day for efficacy measures and baseline characteristics, as well as efficacy durations.

The study day is calculated as below:

- Assessment Date = Missing → Study Day = Missing
- Assessment Date < Reference Date → Study Day = Assessment Date Ref Date
- Assessment Date  $\geq$  Reference Date  $\rightarrow$  Study Day = Assessment Date Ref Date + 1

#### 6.2.7. Assessment Window

Unscheduled and withdrawal visit data will be slotted into a target visit based on visit window defined in the table below. If there are multiple assessments within the same window, the closest one to the target day will be taken in the slotting. If multiple records are equally close to the target day, then the later record will be utilized. For post-baseline records collected outside the analysis visit window, a blank analysis visit label will be assigned.

| Analysis Set / | Parameter (if | Target | Analysis Window | | Analysis |
|---|---|---|---|---|---|
| Domain | applicable) | | Beginning | Ending | Timepoint |
| | | | Timepoint | Timepoint | |
| All | All | Day 3 | Day 2 | Day 5 | On-therapy |
| All | All | Day 12 | Day 9 | Day 16 | Test-of-Cure |
| All | All | Day 28 | Day 21 | Day 31 | Follow-up |

The procedure of the analysis visit assignment is as follows.

- 1. Calculate the analysis days for planned visit, unscheduled visit, and early withdrawal visit with non-missing outcome if applicable. The calculation of the analysis days is provided in Section 6.2.6.
- 2. Slot the visits to each of analysis timepoint according to the above table.
  - a. If there are multiple assessments within the same windows, the closest one to the target day will be taken in the slotting.
  - b. If multiple records are equally close to the target day, then the later record will be utilized using the sequence number in SDTM dataset.
  - c. For post-baseline records collected outside the analysis visit window, a blank analysis visit label will be assigned. Such assessments will not be included in any of the by visit summaries. Descriptive summaries that are shown for "any assessment post baseline" e.g. maximum/minimum/ worst case post baseline, will use all assessments irrespective of whether they fall in an analysis visit window.

# 6.2.8. Multiple measurements at One Analysis Time Point

Not applicable.

# 6.2.9. Handling of Partial Dates

| Element | Reporting Detail | |
|---|---|---|
| General | <ul> <li>Partial dates will</li> <li>However, where variables for sor for 'slotting' data</li> <li>Imputed partial of (e.g., time to one time since diagnocontact date in contact date in contact.</li> </ul> | in the displayed the captainst in participant nearly displayed |
| Adverse Events | conventions: | AE recorded in the CRF will be imputed using the following |
| | Missing start time (AChE-I only) | Midnight 0:00:00 will be used for AEs with missing start time to determine if it's AChE-I. |
| Concomitant Medications/Medical History | Partial dates for using the following that day | any concomitant medications recorded in the CRF will be imputed ng convention: If study intervention start date is missing (i.e. participant did not |
| | | start study intervention), then set start date = 1st of month. Else if study intervention start date is not missing: If month and year of start date = month and year of study intervention start date, then If stop date contains a full date and stop date is earlier than study intervention start date, then set start date= 1st of month. Else set start date = study intervention start date. Else set start date = 1st of month. |
| | Missing start day and month | If study intervention start date is missing (i.e. participant did not start study intervention), then set start date = January 1. Else if study intervention start date is not missing: If year of start date = year of study intervention start date, then If stop date contains a full date and stop date is earlier than study intervention start date, then set start date = January 1. Else set start date = study. intervention start date. Else set start date = January 1. |
| | Missing end day | A '28/29/30/31' will be used for the day (dependent on the month and year). |
| | Missing end day and month | A '31' will be used for the day and 'Dec' will be used for the month. |

| Element | Reporting Detail | |
|---|---|---|
| | Completely missing | No imputation |
| | start/end date | |
| Age | Age is derived using the date of first dose. When first dose date is missing, the informed consent date is used. Only year of birth is collected so Day and Month of birth are imputed | |
| | as 30 June. Formula for deriving age is the integer component of: | |
| | <ul> <li>(First Dose Date</li> </ul> | - 30 Jun of collected birth year + 1) / 365.25 |

# 6.2.10. Qualifying Uropathogen Algorithm

# **Qualifying Uropathogen Decision Tree: Single Uropathogen**



### **Qualifying Uropathogen Decision Tree: 2 Uropathogens**



Note: Since *Enterococcus* spp., beta-hemolytic streptococci, *Gardnerella vaginalis* and *Aerococcus urinae* must be present in pure culture to be considered a uropathogen, the 2 or  $\geq$ 3 uropathogens trees do not apply to these organisms.

#### **Qualifying Uropathogen Decision Tree: >= 3 Uropathogens**



Note: Since *Enterococcus* spp., beta-hemolytic streptococci, *Gardnerella vaginalis* and *Aerococcus urinae* must be present in pure culture to be considered a uropathogen, the 2 or  $\geq$ 3 uropathogens trees do not apply to these organisms.

### 6.2.11. Uropathogen Phenotype Algorithm

### **ESBL. Decision Tree:**



Note: ESBL not determined for other Gram-negative organisms.

## **Methicillin\* Decision Tree:**



\*Cefoxitin is tested as a surrogate test for oxacillin to determine methicillin susceptibility/resistance. Methicillin-(oxacillin) resistant staphylococci are resistant to all currently available beta-lactams, cephalosporin and carbapenem antimicrobial agents, with the exception of ceftaroline.

### **Multidrug Resistance (MDR):**

Definition 1: A uropathogen will be regarded as multidrug-resistant if the uropathogen is resistant to  $\geq$ = 1 drugs in each class among  $\geq$ = 2 antimicrobial classes ( $\beta$ -lactam, Fluoroquinolone, Fosfomycin and Aminoglycoside). This definition will be used for micro-ITT MDR Population.

Definition 2: A uropathogen will be regarded as multidrug-resistant (3 or more) if the uropathogen is resistance to  $\ge 1$  drugs in each class among  $\ge 3$  antimicrobial classes ( $\beta$ -lactam, Fluoroquinolone, Fosfomycin and Aminoglycoside). This phenotype will be included in the subgroup analyses.

Below is the table of antimicrobial classes, susceptibility test and the guideline of susceptibility interpretation for the MDR definitions above.

| Antimicrobial class | <u>Antimicrobial</u> | Susceptibility test | Guideline |
|---|---|---|---|
| | | (MSMETHOD) | (MSSCAT) |
| Beta-lactam | Ampicillin | Micro Broth Dilution | CLSI |
| | Mecillinam | Disk diffusion | CLSI |
| | Penicillin | Disk diffusion | CLSI |
| | Amoxicillin/clavulanic acid | Micro Broth Dilution | CLSI |
| | Ceftolozane/tazobactam | Micro Broth Dilution | CLSI |
| | Ceftazidime/avibactam | Micro Broth Dilution | CLSI |
| | Piperacillin/tazobactam | Micro Broth Dilution | CLSI |
| | Cefazolin | Micro Broth Dilution | CLSI |
| | Ceftriaxone | Micro Broth Dilution | CLSI |
| | Cefadroxil | Disk diffusion | EUCAST |
| | Cefoxitin | Disk diffusion | CLSI |
| | Meropenem | Micro Broth Dilution | CLSI |
| | Faropenem | Disk diffusion | [Fuchs, 1995] |
| Aminoglycoside | Amikacin | Micro Broth Dilution | CLSI |
| | Gentamicin | Micro Broth Dilution | CLSI |
| Fluoroquinolone | Ciprofloxacin | Micro Broth Dilution | CLSI |
| | Levofloxacin | Micro Broth Dilution | CLSI |
| Fosfomycin | Fosfomycin | Agar dilution | CLSI |

### **List of Antimicrobials Being Tested**

| Antimicrobial Class | Sub-class | Antimicrobial |
|---------------------|----------------------|-----------------------------|
| β-lactam | Penicillin | Ampicillin |
| | | Mecillinam |
| | | Penicillin |
| | β-lactam combination | Amoxicillin/clavulanic acid |
| | | Ceftolozane/tazobactam |

| Antimicrobial Class | Sub-class | Antimicrobial |
|---|---|---|
| | | Ceftazidime/avibactam |
| | | Piperacillin/tazobactam |
| | Cephalosporin | Cefazolin |
| | | Ceftriaxone |
| | | Cefotaxime |
| | | Ceftazidime |
| | | Cefpodoxime |
| | | Cefoxitin |
| | | Cefadroxil |
| | | Cefoxitin |
| | Carbapenem/Penem | Meropenem |
| | | Faropenem |
| | Monobactam | Aztrenam |
| Fluoroquinolone | | Ciprofloxacin |
| | | Levofloxacin |
| Fosfomycin | | Fosfomycin |
| Aminoglycoside | | Amikacin |
| | | Gentamicin |
| Folate pathway Antagonist | | Trimethoprim-sulfamethoxazole |
| | | Trimethoprim |
| | | Sulfisoxazole |
| Nitrofuran | | Nitrofurantoin |
| Glycopeptide | | Vancomycin |
| Nitroxoline | | Nitroxoline |

# **Antimicrobial-Resistant Phenotypes:**

| Antimicrobial class | Antimicrobial | Drug<br>relevant to<br>Gram-<br>negatives | Drug<br>relevant to<br>Gram-<br>positives | Resistant<br>phenotype to<br>be reported by<br>GCL if<br>interpretation is<br>resistant* |
|---|---|---|---|---|
| Penicillin | Ampicillin | X | Χ | AMP-R |
| | Mecillinam | Х | | MEC-R |
| | Penicillin | | X | PEN-R |
| B-lactam combination | Amoxicillin/clavulanic acid | Х | | AUG-R |
| | Ceftolozane/tazobactam | Х | | C/T-R |
| | Ceftazidime/avibactam | Х | | CZA-R |
| | Piperacillin/tazobactam | Х | | P/T-R |
| Cephalosporin | Cefazolin | Х | | FAZ-R |
| | Ceftriaxone | Х | | AXO-R |
| | Cefadroxil | Х | | CFR-R |
| | Cefoxitin** | | Х | See methicillin resistance tree |

| Antimicrobial class | Antimicrobial | Drug<br>relevant to<br>Gram-<br>negatives | Drug<br>relevant to<br>Gram-<br>positives | Resistant phenotype to be reported by GCL if interpretation is resistant* |
|---|---|---|---|---|
| Carbapenem/Penem | Meropenem | Х | | MERO-R |
| · | Faropenem | Х | Х | FPM-R |
| Aminoglycoside | Amikacin | Х | | AMI-R |
| | Gentamicin | Х | | GEN-R |
| Folate Pathway | Trimethoprim-sulfamethoxazole | Х | Х | SXT-R |
| Antagonist | Trimethoprim | Х | Х | TMP-R |
| | Sulfisoxazole | Х | Х | SFX-R |
| Fluoroquinolone | Ciprofloxacin | Х | Х | CIP-R |
| | Levofloxacin | Х | Х | LEVO-R |
| Nitrofuran | Nitrofurantoin | Χ | Х | NIT-R |
| Glycopeptide | Vancomycin | | Х | VAN-R |
| Fosfomycin | Fosfomycin | Χ | Х | FOF-R |
| Nitroxoline | Nitroxoline | Χ | Χ | NOX-R |

<sup>\*</sup>Resistant phenotype based on CLSI M100 interpretations with the exception of nitroxoline and cefadroxil which are based on EUCAST interpretations and faropenem which is based on [Fuchs, 1995].

### 6.2.12. Trademarks

| Trademarks of the [GlaxoSmithKline / ViiV<br>Healthcare] Group of Companies |
|---|
| ADVAIR |

| Trademarks not owned by the [GlaxoSmithKline / ViiV Healthcare] Group of Companies |
|---|
| NONMEM |
| SAS |
| WinNonlin |

<sup>\*\*</sup> Surrogate test for oxacillin to determine methicillin susceptibility/resistance. R=resistant

### 7. REFERENCES

Crowe B, Brueckner A, Beasley C, Kulkarni P. Current Practices, Challenges, and Statistical Issues With Product Safety Labeling 2013;5(3): 180-193. *Statistics in Biopharmaceutical Research.* 2013;5(3):180-193.

Fuchs PC, Barry AL, Sewell DL. Antibacterial activity of WY-49605 compared with those of six other oral agents and selection of disk content for disk diffusion susceptibility testing. *Antimicrob Agents Chemother*. 1995;39:1472-9.

SAS Institute Inc. SAS/STAT User's Guide. Version 15.1 ed. Cary, NC:SAS; 2018.

Schmidli HS, Gsteiger S, Roychoudhury S, O'Hagan A, Spiegelhalter D, Neuenschwander B. Robust meta-analytic-predictive priors in clinical trials with historical control information. *Biometrics*. 2014;70:1023-1032.